CLINICAL TRIAL: NCT00328627
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Determine the Efficacy and Safety of the Combination of SYR-322 (SYR110322) and Pioglitazone HCl (ACTOS®), in Subjects With Type 2 Diabetes
Brief Title: Efficacy and Safety of Alogliptin Combined With Pioglitazone in Treating Subjects With Type 2 Diabetes Mellitus.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-05-TL-322OPI-001; 2006-000694-30 (EudraCT Number); U1111-1113-8587 (Registry Identifier: WHO)
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus, Type 2; Drug Therapy; Diabetes Mellitus, Non Insulin Dependent; Glucose Intolerance; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Hyperglycemia | interventions — alogliptin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- Placebo (Placebo Comparator): Alogliptin placebo-matching tablets, orally, once daily and pioglitazone placebo-matching tablets, orally, once daily for up to 26 weeks.
  Interventions: Drug: Alogliptin placebo; Drug: Pioglitazone placebo
- Alogliptin 12.5 + Placebo (Experimental): Alogliptin 12.5 mg, tablets, orally, once daily and pioglitazone placebo-matching tablets, orally, once daily for up to 26 weeks.
  Interventions: Drug: Alogliptin; Drug: Pioglitazone placebo
- Alogliptin 25 + Placebo (Experimental): Alogliptin 25 mg, tablets, orally, once daily and pioglitazone placebo-matching tablets, orally, once daily for up to 26 weeks.
  Interventions: Drug: Alogliptin; Drug: Pioglitazone placebo
- Placebo + Pioglitazone 15 (Active Comparator): Alogliptin placebo-matching tablets, orally, once daily and pioglitazone 15 mg, tablets, orally, once daily for up to 26 weeks.
  Interventions: Drug: Pioglitazone
- Alogliptin 12.5 + Pioglitazone 15 (Experimental): Alogliptin 12.5 mg, tablets, orally, once daily and pioglitazone 15 mg, tablets, orally, once daily for up to 26 weeks.
  Interventions: Drug: Alogliptin; Drug: Pioglitazone
- Alogliptin 25 + Pioglitazone 15 (Experimental): Alogliptin 25 mg, tablets, orally, once daily and pioglitazone 15 mg, tablets, orally, once daily for up to 26 weeks.
  Interventions: Drug: Alogliptin; Drug: Pioglitazone
- Placebo + Pioglitazone 30 (Active Comparator): Alogliptin placebo-matching tablets, orally, once daily and pioglitazone 30 mg, tablets, orally, once daily for up to 26 weeks.
  Interventions: Drug: Alogliptin placebo; Drug: Pioglitazone
- Alogliptin 12.5 + Pioglitazone 30 (Experimental): Alogliptin 12.5 mg, tablets, orally, once daily and pioglitazone 30 mg, tablets, orally, once daily for up to 26 weeks.
  Interventions: Drug: Alogliptin; Drug: Pioglitazone
- Alogliptin 25 + Pioglitazone 30 (Experimental): Alogliptin 25 mg, tablets, orally, once daily and pioglitazone 30 mg, tablets, orally, once daily for up to 26 weeks.
  Interventions: Drug: Alogliptin; Drug: Pioglitazone
- Placebo + Pioglitazone 45 (Active Comparator): Alogliptin placebo-matching tablets, orally, once daily and pioglitazone 45 mg, tablets, orally, once daily for up to 26 weeks.
  Interventions: Drug: Alogliptin placebo; Drug: Pioglitazone
- Alogliptin 12.5 + Pioglitazone 45 (Experimental): Alogliptin 12.5 mg, tablets, orally, once daily and pioglitazone 45 mg, tablets, orally, once daily for up to 26 weeks.
  Interventions: Drug: Alogliptin; Drug: Pioglitazone
- Alogliptin 25 + Pioglitazone 45 (Experimental): Alogliptin 25 mg, tablets, orally, once daily and pioglitazone 45 mg, tablets, orally, once daily for up to 26 weeks.
  Interventions: Drug: Alogliptin; Drug: Pioglitazone

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets.
  Other Names: SYR-322
  Arms: Alogliptin 12.5 + Pioglitazone 15; Alogliptin 12.5 + Pioglitazone 30; Alogliptin 12.5 + Pioglitazone 45; Alogliptin 12.5 + Placebo; Alogliptin 25 + Pioglitazone 15; Alogliptin 25 + Pioglitazone 30; Alogliptin 25 + Pioglitazone 45; Alogliptin 25 + Placebo
Drug: Alogliptin placebo — Alogliptin placebo-matching tablets.
  Arms: Placebo; Placebo + Pioglitazone 30; Placebo + Pioglitazone 45
Drug: Pioglitazone — Pioglitazone tablets.
  Other Names: ACTOS®
  Arms: Alogliptin 12.5 + Pioglitazone 15; Alogliptin 12.5 + Pioglitazone 30; Alogliptin 12.5 + Pioglitazone 45; Alogliptin 25 + Pioglitazone 15; Alogliptin 25 + Pioglitazone 30; Alogliptin 25 + Pioglitazone 45; Placebo + Pioglitazone 15; Placebo + Pioglitazone 30; Placebo + Pioglitazone 45
Drug: Pioglitazone placebo — Pioglitazone placebo-matching tablets.
  Arms: Alogliptin 12.5 + Placebo; Alogliptin 25 + Placebo; Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of alogliptin, once daily (QD), taken in combination with pioglitazone in adults with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Over the past 30 years, the prevalence of diabetes has increased dramatically throughout the world due to population growth, aging, urbanization, increasing obesity, and physical inactivity. The total number of people with type 2 diabetes mellitus is projected to rise from 171 million in 2000 to 366 million in 2030. The incidence of type 2 diabetes mellitus in the United States alone is expected to increase from approximately 17 to 30.3 million by the year 2030. Type 2 diabetes mellitus is associated with a number of long-term microvascular and macrovascular complications associated with a reduced quality of life and increased morbidity and mortality. It is anticipated that the increasing incidence of type 2 diabetes mellitus will place an ever-increasing burden on families, increase national expenditures for health care services, and decrease worker productivity.

Current pharmacologic interventions for type 2 diabetes mellitus include a diverse range of antidiabetic medications with different mechanisms of action including insulin and insulin analogues, sulfonylureas, metformin, meglitinides, thiazolidinediones, inhibitors of alpha-glucosidase, analogs of glucagon-like peptide-1 and synthetic analogues of human amylin. Despite the variety of medications, many have clinically important or potentially life-threatening side effects, restricted use in many subpopulations, concerns with long-term tolerability, and challenges related to compliance due to side effects and route of administration. All of these reasons contribute to the difficulties patients have achieving the target glycosylated hemoglobin level less than 7%.

SYR-322 (alogliptin) is a selective, orally available inhibitor of the dipeptidyl peptidase-4 enzyme. Dipeptidyl peptidase-4 enzyme is thought to be primarily responsible for the in vivo degradation of 2 peptide hormones released in response to nutrient ingestion, namely glucagon-like peptide-1 and glucose-dependent insulinotropic peptide. Both peptides exert important effects on islet beta cells to stimulate glucose-dependent insulin secretion as well as regulating beta cell proliferation and cytoprotection. Glucagon-like peptide-1, but not glucose-dependent insulinotropic peptide, inhibits gastric emptying, glucagon secretion, and food intake. Glucose-dependent insulinotropic peptide has been shown to enhance insulin secretion by direct interaction with a glucose-dependent insulinotropic peptide -specific receptor on islet beta cells. The glucose-lowering actions of glucagon-like peptide-1, but not glucose-dependent insulinotropic peptide, are preserved in patients with type 2 diabetes mellitus.

Pioglitazone (ACTOS®) is a thiazolidinedione developed by Takeda Chemical Industries, Ltd. (Osaka, Japan) that is approved for the treatment of type 2 diabetes mellitus. Pioglitazone is a selective peroxisome proliferator-activated receptor-gamma agonist that decreases insulin resistance in the periphery and liver resulting in increased insulin-dependent glucose disposal and decreased hepatic glucose output.

Given the complementary mechanisms of action of alogliptin (stimulation of insulin secretion) and pioglitazone (enhancement of insulin sensitivity), the goal of this study is to evaluate the efficacy of the combination of alogliptin with pioglitazone in patients who are inadequately controlled on metformin. Study participation is anticipated to be approximately 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with a historical diagnosis of type 2 diabetes mellitus who were treated with metformin greater than or equal to 1500 mg alone but were experiencing inadequate glycemic control.
* A stable dose of metformin of greater than or equal to 1500 mg or maximum tolerated dose.
* No treatment with antidiabetic agents other than metformin within the 2 months prior to Screening.
* A body mass index greater than or equal to 23 kg/m^2 and less than or equal to 45 kg/m^2.
* Fasting C-peptide greater than or equal to 0.8 ng/mL.
* Regular use of other, non-excluded medications was allowed if a stable dose had been established for at least 4 weeks prior to Screening.
* Systolic blood pressure less than or equal to 160 mmHg and diastolic pressure less than or equal to 100 mmHg.
* Hemoglobin greater than or equal to 12 g/dL for men and greater than or equal to 10 g/dL for women.
* Alanine aminotransferase less than or equal to 2.5 times the upper limit of normal.
* Serum creatinine less than 1.5 mg/dL for men and less than 1.4 mg/dL for women.
* Thyroid-stimulating hormone level less than or equal to the upper limit of the normal range and the subject was clinically euthyroid.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Able and willing to monitor their own blood glucose concentrations with a home glucose monitor.
* No major illness or debility that in the investigator's opinion prohibited the patient from completing the study.

Exclusion Criteria:

* Urine albumin/creatinine ratio greater than 113 mg/mmol at Screening.
* A history of cancer, other than squamous cell or basal cell carcinoma of the skin, that had not been in full remission for at least 5 years prior to Screening.
* A history of laser treatment for proliferative diabetic retinopathy within 6 months prior to Screening.
* A history of treated diabetic gastroparesis.
* New York Heart Association Class III or IV heart failure regardless of therapy.
* History of coronary angioplasty, coronary stent placement, coronary bypass surgery, or myocardial infarction within the 6 months prior to Screening.
* History of any hemoglobinopathy.
* History of infection with hepatitis B, hepatitis C or human immunodeficiency virus.
* History of a psychiatric disorder that could have affected the patient's ability to participate in the study.
* History of angioedema in association with use of angiotensin-converting enzyme inhibitors or angiotensin-II receptor inhibitors.
* A history of alcohol or substance abuse within 2 years prior to Screening.
* Receipt of any investigational drug within 30 days prior to Screening or a history of receipt of an investigational antidiabetic drug within 3 months prior to Screening.
* Previous participation in an investigational study of alogliptin.
* Hypersensitive to pioglitazone, alogliptin, or other excipients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1554 (Actual)
Dates: Start 2006-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP Biological Sciences, Study Director — Takeda
Locations (90):
- United States (72):
  - Birmingham, Alabama
  - Columbiana, Alabama
  - Huntsville, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Searcy, Arkansas
  - Sherwood, Arkansas
  - Burbank, California
  - Foothill Ranch, California
  - Irvine, California
  - Sacramento, California
  - San Diego, California
  - Temecula, California
  - Tustin, California
  - Colorado Springs, Colorado
  - Washington D.C., District of Columbia
  - Hollywood, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - Sarasota, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Roswell, Georgia
  - Savannah, Georgia
  - Warner Robins, Georgia
  - Chicago, Illinois
  - Peoria, Illinois
  - Lafayette, Indiana
  - South Bend, Indiana
  - Waterloo, Iowa
  - Munfordville, Kentucky
  - Baton Rouge, Louisiana
  - Marrero, Louisiana
  - Elkridge, Maryland
  - Prince Frederick, Maryland
  - Towson, Maryland
  - Marlborough, Massachusetts
  - Ann Arbor, Michigan
  - Cadillac, Michigan
  - Detroit, Michigan
  - Livonia, Michigan
  - Kansas City, Missouri
  - North Las Vegas, Nevada
  - Blackwood, New Jersey
  - Trenton, New Jersey
  - New York, New York
  - Charlotte, North Carolina
  - Statesville, North Carolina
  - Gallipolis, Ohio
  - Marion, Ohio
  - Clinton, Oklahoma
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Allentown, Pennsylvania
  - Altoona, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Alcoa, Tennessee
  - Milan, Tennessee
  - Morristown, Tennessee
  - Arlington, Texas
  - Carrollton, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
- Multiple Cities, Australia
- Multiple Cities, Brazil
- Multiple Cities, Bulgaria
- Multiple Cities, Chile
- Multiple Cities, Croatia
- Multiple Cities, Estonia
- Multiple Cities, Guatemala
- Multiple Cities, India
- Multiple Cities, Israel
- Multiple Cities, Latvia
- Multiple Cities, Mexico
- Multiple Cities, New Zealand
- Multiple Cities, Peru
- Multiple Cities, Romania
- Multiple Cities, Russia
- Multiple Cities, Serbia
- Multiple Cities, South Africa
- Multiple Cities, Ukraine

REFERENCES:
- [Result] DeFronzo RA, Burant CF, Fleck P, Wilson C, Mekki Q, Pratley RE. Efficacy and tolerability of the DPP-4 inhibitor alogliptin combined with pioglitazone, in metformin-treated patients with type 2 diabetes. J Clin Endocrinol Metab. 2012 May;97(5):1615-22. doi: 10.1210/jc.2011-2243. Epub 2012 Mar 14. PMID 22419732
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 327 investigative sites in 20 countries from 31 May 2006 to 17 March 2008.
Pre-assignment Details: Participants with a diagnosis of type 2 diabetes who were inadequately controlled on a regimen of metformin alone were equally randomized to 1 of 12 double-blind treatment groups.
Period: Overall Study
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Started | 129 | 128 | 129 | 130 | 130 | 130 | 129 | 130 | 130 | 129 | 130 | 130
Safety Set | 129 (All patients who took at least 1 dose of double-blind study drug.) | 128 | 129 | 129 | 130 | 130 | 129 | 130 | 130 | 129 | 130 | 130
Completed | 70 | 97 | 101 | 93 | 115 | 110 | 94 | 116 | 113 | 97 | 112 | 114
Not Completed | 59 | 31 | 28 | 37 | 15 | 20 | 35 | 14 | 17 | 32 | 18 | 16
Not completed — Hyperglycemic Rescue | 41 | 18 | 16 | 13 | 6 | 5 | 19 | 6 | 6 | 11 | 3 | 2
Not completed — Adverse Event | 3 | 1 | 2 | 3 | 1 | 2 | 1 | 2 | 0 | 7 | 5 | 4
Not completed — Protocol Violation | 2 | 2 | 2 | 8 | 5 | 5 | 6 | 2 | 1 | 4 | 6 | 2
Not completed — Lost to Follow-up | 4 | 2 | 2 | 4 | 0 | 2 | 3 | 0 | 3 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 4 | 5 | 6 | 2 | 5 | 4 | 4 | 4 | 5 | 2 | 7
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 3 | 1 | 2 | 1 | 1 | 1 | 0 | 3 | 2 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45 | Total
Number analyzed (Participants) | 129 | 128 | 129 | 130 | 130 | 130 | 129 | 130 | 130 | 129 | 130 | 130 | 1554
Age Continuous [Mean (Standard Deviation); unit: years] | 55.2 (9.89) | 53.1 (9.59) | 53.7 (9.31) | 54.1 (9.54) | 53.6 (9.91) | 54.9 (9.18) | 56.1 (9.43) | 55.0 (9.07) | 54.4 (9.69) | 54.5 (9.70) | 54.0 (9.82) | 54.2 (8.86) | 54.4 (9.50)
Age, Customized [Number; unit: participants]
  <65 years | 106 | 116 | 112 | 113 | 109 | 112 | 101 | 111 | 107 | 112 | 111 | 112 | 1322
  ≥65 years | 23 | 12 | 17 | 17 | 21 | 18 | 28 | 19 | 23 | 17 | 19 | 18 | 232
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 61 | 79 | 69 | 70 | 69 | 66 | 76 | 75 | 76 | 70 | 78 | 857
  Male | 61 | 67 | 50 | 61 | 60 | 61 | 63 | 54 | 55 | 53 | 60 | 52 | 697
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63 | 60 | 63 | 63 | 55 | 57 | 67 | 66 | 62 | 61 | 63 | 65 | 745
  Not Hispanic or Latino | 66 | 68 | 66 | 67 | 75 | 73 | 62 | 64 | 68 | 68 | 67 | 65 | 809
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 5
  Asian | 5 | 14 | 15 | 11 | 9 | 7 | 10 | 5 | 12 | 12 | 8 | 12 | 120
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 6 | 5 | 8 | 4 | 3 | 6 | 2 | 5 | 9 | 9 | 3 | 68
  White | 93 | 89 | 80 | 85 | 95 | 96 | 96 | 107 | 85 | 85 | 92 | 93 | 1096
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 23 | 19 | 29 | 26 | 20 | 22 | 17 | 15 | 28 | 23 | 21 | 22 | 265
Weight [Mean (Standard Deviation); unit: kg] | 83.38 (18.378) | 84.63 (19.378) | 83.25 (18.326) | 84.68 (18.634) | 85.95 (18.498) | 82.90 (16.570) | 85.86 (20.347) | 83.68 (18.340) | 85.77 (18.844) | 82.10 (17.019) | 85.01 (18.536) | 82.79 (18.768) | 84.17 (18.470)
Height [Mean (Standard Deviation); unit: cm] | 164.48 (10.157) | 164.61 (10.614) | 162.38 (9.790) | 164.25 (11.007) | 164.59 (10.841) | 163.74 (10.456) | 164.59 (9.724) | 163.63 (11.036) | 163.64 (9.548) | 163.14 (10.961) | 163.82 (10.708) | 163.73 (11.432) | 163.88 (10.522)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.59 (4.808) | 30.96 (5.133) | 31.48 (5.733) | 31.25 (5.280) | 31.53 (4.979) | 30.78 (4.723) | 31.41 (5.391) | 31.09 (5.054) | 31.86 (5.585) | 30.69 (4.721) | 31.51 (5.206) | 30.62 (4.751) | 31.15 (5.122)
Diabetes Duration [Mean (Standard Deviation); unit: years] | 6.01 (4.958) | 6.17 (5.614) | 5.55 (4.879) | 5.70 (4.767) | 6.08 (5.485) | 6.86 (5.489) | 7.63 (7.069) | 5.81 (5.054) | 6.63 (6.005) | 5.68 (4.232) | 6.59 (5.273) | 6.22 (5.014) | 6.24 (5.375)
Baseline metformin dose [Mean (Standard Deviation); unit: mg] | 1936.8 (428.41) | 1902.0 (450.17) | 1851.2 (413.85) | 1892.6 (410.70) | 1909.6 (418.98) | 1880.0 (413.65) | 1853.5 (435.72) | 1822.3 (444.22) | 1867.1 (455.48) | 1918.6 (417.91) | 1919.6 (421.22) | 1884.6 (439.47) | 1886.5 (429.08)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 26 in Glycosylated Hemoglobin (HbA1c) (Grouped Analysis)
Description: The change from Baseline to Week 26 in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound).
  The primary analysis compared the groupings (combinations of individual treatment groups) of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone (Pioglitazone Alone).
Time Frame: Baseline and Week 26
Population: Full analysis set where Baseline and at least 1 postbaseline assessment were available. Last observation carried forward imputation was utilized.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Groups:
- Pioglitazone Alone: Alogliptin placebo plus all active pioglitazone groups (15, 30, and 45 mg).
  This combination group includes participants from the following three treatment arms:
  1. Placebo + Pioglitazone 15 mg
  2. Placebo + Pioglitazone 30 mg
  3. Placebo + Pioglitazone 45 mg
- Alogliptin 12.5 + Pioglitazone: Alogliptin 12.5 mg plus all active pioglitazone (15, 30, and 45 mg).
  This combination group includes participants from the following three treatment arms:
  1. Alogliptin 12.5 mg + Pioglitazone 15 mg
  2. Alogliptin 12.5 mg + Pioglitazone 30 mg
  3. Alogliptin 12.5 mg + Pioglitazone 45 mg
- Alogliptin 25 + Pioglitazone: Alogliptin 25 mg plus all active pioglitazone (15, 30, and 45 mg).
  This combination group includes participants from the following three treatment arms:
  1. Alogliptin 25 mg + Pioglitazone 15 mg
  2. Alogliptin 25 mg + Pioglitazone 30 mg
  3. Alogliptin 25 mg + Pioglitazone 45 mg
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 376 | 385 | 377
percentage of glycosylated hemoglobin | -0.89 (0.046) | -1.43 (0.046) | -1.42 (0.046)
Statistical Analysis 1: Comparison: Pioglitazone Alone vs Alogliptin 12.5 + Pioglitazone; The null hypothesis was that the doses of alogliptin do not have any additive effect on glycemic control (HbA1c) in addition to the effect produced by pioglitazone alone. The alternative hypothesis was that at least the higher dose of alogliptin would have an additive effect on glycemic control (HbA1c) in addition to the effect produced by pioglitazone alone; Test type: Superiority or Other; p < 0.001, ANCOVA — For the primary analysis, the overall average HbA1c response of the Alogliptin/pioglitazone combination groups was compared with that of the pioglitazone alone groups at the 2-sided 0.05 significance level with no adjustment for multiple comparisons; ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline HbA1c as continuous covariates; LS Mean Difference = -0.54, 95% CI 2-sided [-0.67 to -0.41]
Statistical Analysis 2: Comparison: Pioglitazone Alone vs Alogliptin 25 + Pioglitazone; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.53, 95% CI 2-sided [-0.66 to -0.41]

2. Secondary Outcome: Change From Baseline in HbA1c Over Time (Grouped Analysis)
Description: The change from Baseline to Weeks 4, 8, 12, 16 and 20 in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound).
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an analysis of covariance (ANCOVA) model with treatment and geographic region as class variables, and baseline metformin dose and HbA1c as continuous covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16 and 20.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Groups:
- Pioglitazone Alone: Alogliptin placebo plus all active pioglitazone groups (15, 30, and 45 mg).
- Alogliptin 12.5 + Pioglitazone: Alogliptin 12.5 mg plus all active pioglitazone (15, 30, and 45 mg).
- Alogliptin 25 + Pioglitazone: Alogliptin 25 mg plus all active pioglitazone (15, 30, and 45 mg).
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
percentage of glycosylated hemoglobin
  Week 4 (n=345, 359, 346) | -0.32 (0.023) | -0.57 (0.023) | -0.61 (0.023)
  Week 8 (n=376, 385, 377) | -0.61 (0.034) | -1.06 (0.033) | -1.09 (0.034)
  Week 12 (n=376, 385, 377) | -0.81 (0.039) | -1.29 (0.039) | -1.38 (0.039)
  Week 16 (n=376, 385, 377) | -0.92 (0.041) | -1.44 (0.041) | -1.49 (0.041)
  Week 20 (n=376, 385, 377) | -0.92 (0.043) | -1.46 (0.042) | -1.51 (0.043)

3. Secondary Outcome: Change From Baseline to Week 4 in HbA1c
Description: The change from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) at week 4. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline HbA1c as continuous covariates.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 120 | 114 | 110 | 114 | 120 | 116 | 116 | 122 | 118 | 115 | 117 | 112
percentage of glycosylated hemoglobin | -0.22 (0.039) | -0.46 (0.040) | -0.51 (0.041) | -0.32 (0.040) | -0.53 (0.039) | -0.61 (0.040) | -0.24 (0.040) | -0.60 (0.039) | -0.60 (0.039) | -0.40 (0.040) | -0.58 (0.040) | -0.63 (0.040)

4. Secondary Outcome: Change From Baseline to Week 8 in HbA1c
Description: The change from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) at week 8. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline HbA1c as continuous covariates.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Groups:
- Alogliptin 12.5 mg + Pioglitazone 30 mg: Alogliptin 12.5 mg, tablets, orally, once daily and pioglitazone 30 mg, tablets, orally, once daily for up to 26 weeks.
- Placebo + Pioglitazone 45 mg: Alogliptin placebo-matching tablets, orally, once daily and pioglitazone 45 mg, tablets, orally, once daily for up to 26 weeks.
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 mg + Pioglitazone 30 mg | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 mg | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 126 | 122 | 123 | 127 | 130 | 127 | 123 | 128 | 124 | 126 | 127 | 126
percentage of glycosylated hemoglobin | -0.30 (0.058) | -0.75 (0.059) | -0.80 (0.059) | -0.50 (0.058) | -1.01 (0.058) | -1.04 (0.058) | -0.57 (0.059) | -1.05 (0.058) | -1.02 (0.059) | -0.76 (0.058) | -1.11 (0.058) | -1.20 (0.058)

5. Secondary Outcome: Change From Baseline to Week 12 in HbA1c
Description: The change from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) at week 12.
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline HbA1c as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 mg + Pioglitazone 30 mg | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 mg | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 126 | 122 | 123 | 127 | 130 | 127 | 123 | 128 | 124 | 126 | 127 | 126
percentage of glycosylated hemoglobin | -0.28 (0.067) | -0.84 (0.069) | -0.92 (0.068) | -0.65 (0.067) | -1.24 (0.066) | -1.26 (0.067) | -0.77 (0.068) | -1.29 (0.067) | -1.33 (0.068) | -1.02 (0.067) | -1.34 (0.067) | -1.53 (0.067)

6. Secondary Outcome: Change From Baseline to Week 16 in HbA1c
Description: The change from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) at week 16. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline HbA1c as continuous covariates.
Time Frame: Baseline and Week 16
Population: Full analysis set where Baseline and at least 1 postbaseline assessment were available. Last observation carried forward (LOCF) imputation was utilized.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 mg + Pioglitazone 30 mg | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 mg | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 126 | 122 | 123 | 127 | 130 | 127 | 123 | 128 | 124 | 126 | 127 | 126
percentage of glycosylated hemoglobin | -0.27 (0.071) | -0.82 (0.072) | -1.03 (0.072) | -0.74 (0.071) | -1.36 (0.070) | -1.36 (0.071) | -0.91 (0.072) | -1.42 (0.071) | -1.45 (0.072) | -1.12 (0.071) | -1.53 (0.071) | -1.66 (0.071)

7. Secondary Outcome: Change From Baseline to Week 20 in HbA1c
Description: The change from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) at week 20.
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline HbA1c as continuous covariates.
Time Frame: Baseline and Week 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 mg + Pioglitazone 30 mg | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 mg | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 126 | 122 | 123 | 127 | 130 | 127 | 123 | 128 | 124 | 126 | 127 | 126
percentage of glycosylated hemoglobin | -0.24 (0.074) | -0.75 (0.075) | -0.99 (0.075) | -0.75 (0.074) | -1.39 (0.073) | -1.37 (0.074) | -0.90 (0.075) | -1.43 (0.074) | -1.49 (0.075) | -1.10 (0.074) | -1.57 (0.074) | -1.66 (0.074)

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose Over Time (Grouped Analysis)
Description: The change from Baseline in fasting plasma glucose was assessed at weeks 1, 2, 4, 8, 12, 16, 20 and 26.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline fasting plasma glucose as covariates.
Time Frame: Baseline and Weeks 1, 2, 4, 8, 12, 16, 20 and 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
mg/dL
  Week 1 (n=358, 355, 354) | -4.1 (1.56) | -22.6 (1.57) | -23.1 (1.57)
  Week 2 (n=379, 383, 381) | -11.3 (1.62) | -30.3 (1.61) | -31.6 (1.62)
  Week 4 (n=381, 386, 383) | -19.9 (1.67) | -36.8 (1.66) | -39.8 (1.67)
  Week 8 (n=381, 386, 383) | -27.3 (1.77) | -42.3 (1.76) | -45.2 (1.77)
  Week 12 (n=381, 386, 383) | -30.3 (1.84) | -45.0 (1.83) | -47.6 (1.83)
  Week 16 (n=381, 386, 383) | -27.9 (1.86) | -43.7 (1.85) | -45.4 (1.86)
  Week 20 (n=381, 386, 383) | -28.1 (2.00) | -43.6 (1.99) | -45.0 (1.99)
  Week 26 (n=381, 386, 383) | -28.3 (2.03) | -45.2 (2.02) | -44.2 (2.03)

9. Secondary Outcome: Change From Baseline to Week 1 in Fasting Plasma Glucose
Description: Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline fasting plasma glucose as covariates.
Time Frame: Baseline and Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 123 | 114 | 117 | 120 | 121 | 123 | 117 | 119 | 118 | 121 | 115 | 113
mg/dL | 1.8 (2.67) | -14.5 (2.77) | -18.6 (2.73) | -6.1 (2.70) | -21.3 (2.69) | -20.9 (2.66) | 0.4 (2.73) | -23.2 (2.71) | -23.2 (2.72) | -6.7 (2.69) | -23.2 (2.76) | -25.0 (2.78)

10. Secondary Outcome: Change From Baseline to Week 2 in Fasting Plasma Glucose
Description: as for outcome 9
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 129 | 120 | 125 | 127 | 127 | 129 | 124 | 128 | 126 | 128 | 128 | 126
mg/dL | 4.8 (2.78) | -21.9 (2.88) | -18.9 (2.82) | -10.4 (2.80) | -30.1 (2.80) | -31.7 (2.78) | -4.3 (2.83) | -30.0 (2.79) | -31.3 (2.81) | -19.3 (2.79) | -30.8 (2.79) | -31.7 (2.81)

11. Secondary Outcome: Change From Baseline to Week 4 in Fasting Plasma Glucose
Description: as for outcome 9
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 129 | 122 | 125 | 127 | 129 | 130 | 125 | 129 | 126 | 129 | 128 | 127
mg/dL | 3.8 (2.87) | -20.4 (2.95) | -22.8 (2.92) | -20.2 (2.90) | -35.3 (2.87) | -37.3 (2.86) | -13.4 (2.92) | -37.4 (2.88) | -36.0 (2.91) | -26.1 (2.87) | -37.8 (2.89) | -46.2 (2.89)

12. Secondary Outcome: Change From Baseline to Week 8 in Fasting Plasma Glucose
Description: as for outcome 9
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 129 | 122 | 126 | 127 | 129 | 130 | 125 | 129 | 126 | 129 | 128 | 127
mg/dL | 5.7 (3.05) | -19.5 (3.14) | -19.3 (3.09) | -22.2 (3.07) | -42.3 (3.05) | -39.3 (3.04) | -24.0 (3.10) | -40.5 (3.05) | -44.1 (3.08) | -35.6 (3.05) | -44.0 (3.06) | -52.3 (3.07)

13. Secondary Outcome: Change From Baseline to Week 12 in Fasting Plasma Glucose
Description: as for outcome 9
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 129 | 122 | 126 | 127 | 129 | 130 | 125 | 129 | 126 | 129 | 128 | 127
mg/dL | 3.4 (3.16) | -19.3 (3.25) | -23.3 (3.19) | -23.0 (3.18) | -42.9 (3.16) | -42.5 (3.14) | -26.6 (3.21) | -42.8 (3.16) | -49.0 (3.19) | -41.3 (3.16) | -49.2 (3.17) | -51.4 (3.18)

14. Secondary Outcome: Change From Baseline to Week 16 in Fasting Plasma Glucose
Description: as for outcome 9
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 129 | 122 | 126 | 127 | 129 | 130 | 125 | 129 | 126 | 129 | 128 | 127
mg/dL | 1.4 (3.20) | -16.2 (3.29) | -22.6 (3.24) | -21.2 (3.22) | -41.6 (3.20) | -39.1 (3.19) | -26.3 (3.25) | -41.5 (3.20) | -43.4 (3.24) | -36.3 (3.20) | -47.9 (3.21) | -53.8 (3.22)

15. Secondary Outcome: Change From Baseline to Week 20 in Fasting Plasma Glucose
Description: as for outcome 9
Time Frame: Baseline and Week 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 129 | 122 | 126 | 127 | 129 | 130 | 125 | 129 | 126 | 129 | 128 | 127
mg/dL | 6.7 (3.43) | -8.7 (3.53) | -23.5 (3.48) | -22.4 (3.46) | -43.0 (3.43) | -39.3 (3.42) | -26.3 (3.49) | -41.1 (3.44) | -43.1 (3.47) | -35.7 (3.43) | -46.8 (3.45) | -52.4 (3.46)

16. Secondary Outcome: Change From Baseline to Week 26 in Fasting Plasma Glucose
Description: as for outcome 9
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 129 | 122 | 126 | 127 | 129 | 130 | 125 | 129 | 126 | 129 | 128 | 127
mg/dL | 6.5 (3.50) | -13.2 (3.59) | -18.6 (3.54) | -23.6 (3.52) | -42.0 (3.50) | -38.0 (3.48) | -28.8 (3.55) | -42.2 (3.50) | -41.7 (3.54) | -32.4 (3.49) | -51.3 (3.51) | -52.7 (3.52)

17. Secondary Outcome: Percentage of Participants With Marked Hyperglycemia (Grouped Analysis)
Description: Marked hyperglycemia is defined as fasting plasma glucose greater than or equal to 200 mg/dL (11.10 mmol/L).
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone.
Time Frame: From Week 1 to Week 26
Population: Full analysis set including patients with at least one non-missing fasting plasma glucose result in each treatment group.
Measure: Number; unit: percentage of participants
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 381 | 386 | 384
percentage of participants | 39.4 | 24.6 | 22.1

18. Secondary Outcome: Percentage of Participants With Marked Hyperglycemia
Description: Marked hyperglycemia is defined as fasting plasma glucose greater than or equal to 200 mg/dL (11.10 mmol/L).
Time Frame: From Week 1 to Week 26
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 129 | 122 | 126 | 127 | 129 | 130 | 125 | 129 | 127 | 129 | 128 | 127
percentage of participants | 60.5 | 42.6 | 39.7 | 37.8 | 27.1 | 22.3 | 39.2 | 26.4 | 23.6 | 41.1 | 20.3 | 20.5

19. Secondary Outcome: Percentage of Participants Meeting Rescue Criteria (Grouped Analysis)
Description: Rescue was defined as meeting 1 of the following criteria, confirmed by a 2nd sample drawn within 5 days of the first and analyzed by the central laboratory:
  1. After the Week 1 Visit but prior to the Week 4 Visit: a single fasting plasma glucose ≥300 mg/dL;
  2. From the Week 4 Visit but prior to the Week 8 Visit: a single fasting plasma glucose ≥275 mg/dL;
  3. From the Week 8 Visit but prior to the Week 12 Visit: a single fasting plasma glucose ≥250 mg/dL;
  4. From the Week 12 Visit through the End-of-Treatment Visit: HbA1c ≥8.5% and ≤0.5% reduction in HbA1c as compared with Baseline HbA1c.
Time Frame: From Week 1 to Week 26.
Population: Full analysis set including patients with at least 1 postbaseline visit. This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone.
Measure: Number; unit: percentage of participants
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 376 | 382 | 377
percentage of participants | 11.4 | 3.9 | 3.4

20. Secondary Outcome: Percentage of Participants Meeting Rescue Criteria
Description: as for outcome 19
Time Frame: From Week 1 to Week 26
Population: Full analysis set including patients with at least 1 postbaseline visit.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 124 | 125 | 127 | 129 | 129 | 123 | 126 | 123 | 126 | 127 | 125
percentage of participants | 32.8 | 14.5 | 12.8 | 10.2 | 4.7 | 3.9 | 15.4 | 4.8 | 4.9 | 8.7 | 2.4 | 1.6

21. Secondary Outcome: Percentage of Participants With Glycosylated Hemoglobin ≤ 6.5% (Grouped Analysis)
Description: Clinical response at Week 26 was assessed by the percentage of participants with HbA1c less than or equal to 6.5%.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone.
Time Frame: Week 26
Population: The full analysis set. Patients who did not complete the scheduled Week 26 visit were assessed based on their response at the time of discontinuation.
Measure: Number; unit: percentage of participants
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
percentage of participants | 12.4 | 27.9 | 29.2

22. Secondary Outcome: Percentage of Participants With Glycosylated Hemoglobin ≤ 6.5%
Description: Clinical response at Week 26 was assessed by the percentage of participants with HbA1c less than or equal to 6.5%.
Time Frame: Week 26
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 129 | 128 | 129 | 129 | 130 | 130 | 129 | 130 | 130 | 129 | 130 | 130
percentage of participants | 0.8 | 8.6 | 12.4 | 6.2 | 21.5 | 24.6 | 11.6 | 30.0 | 30.0 | 19.4 | 32.3 | 33.1

23. Secondary Outcome: Percentage of Participants With Glycosylated Hemoglobin ≤ 7.0% (Grouped Analysis)
Description: Clinical response at Week 26 was assessed by the percentage of participants with HbA1c less than or equal to 7%.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone.
Time Frame: Week 26
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
percentage of participants | 30.5 | 54.6 | 55.9

24. Secondary Outcome: Percentage of Participants With Glycosylated Hemoglobin ≤ 7%
Description: Clinical response at Week 26 was assessed by the percentage of participants with HbA1c less than or equal to 7%.
Time Frame: Week 26
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 129 | 128 | 129 | 129 | 130 | 130 | 129 | 130 | 130 | 129 | 130 | 130
percentage of participants | 6.2 | 22.7 | 27.1 | 25.6 | 49.2 | 54.6 | 29.5 | 53.1 | 53.1 | 36.4 | 61.5 | 60.0

25. Secondary Outcome: Percentage of Participants With Glycosylated Hemoglobin ≤ 7.5% (Grouped Analysis)
Description: Clinical response at Week 26 was assessed by the percentage of participants with HbA1c less than or equal to 7.5%.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone.
Time Frame: Week 26
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
percentage of participants | 54.8 | 77.4 | 74.1

26. Secondary Outcome: Percentage of Participants With Glycosylated Hemoglobin ≤ 7.5%
Description: Clinical response at Week 26 was assessed by the percentage of participants with HbA1c less than or equal to 7.5%.
Time Frame: Week 26
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 129 | 128 | 129 | 129 | 130 | 130 | 129 | 130 | 130 | 129 | 130 | 130
percentage of participants | 24.8 | 38.3 | 55.0 | 51.9 | 77.7 | 71.5 | 55.8 | 73.8 | 72.3 | 56.6 | 80.8 | 78.5

27. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin ≥ 0.5% (Grouped Analysis)
Description: Clinical response at Week 26 was assessed by the percentage of participants with a decrease from Baseline in HbA1c of greater than or equal to 0.5%.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone.
Time Frame: Baseline and Week 26
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
percentage of participants | 67.2 | 85.6 | 83.3

28. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin ≥ 0.5%
Description: Clinical response at Week 26 was assessed by the percentage of participants with a decrease from Baseline in HbA1c of greater than or equal to 0.5%.
Time Frame: Baseline and Week 26
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 129 | 128 | 129 | 129 | 130 | 130 | 129 | 130 | 130 | 129 | 130 | 130
percentage of participants | 31.8 | 57.8 | 66.7 | 61.2 | 86.2 | 79.2 | 68.2 | 86.9 | 83.8 | 72.1 | 83.8 | 86.9

29. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin ≥ 1% (Grouped Analysis)
Description: Clinical response at Week 26 was assessed by the percentage of participants with a decrease from Baseline in HbA1c of greater than or equal to 1%.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone.
Time Frame: Baseline and Week 26
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
percentage of participants | 45.7 | 71.8 | 69.5

30. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin ≥ 1%
Description: Clinical response at Week 26 was assessed by the percentage of participants with a decrease from Baseline in HbA1c of greater than or equal to 1%.
Time Frame: Baseline and Week 26
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 129 | 128 | 129 | 129 | 130 | 130 | 129 | 130 | 130 | 129 | 130 | 130
percentage of participants | 16.3 | 33.6 | 47.3 | 36.4 | 69.2 | 66.9 | 46.5 | 73.1 | 69.2 | 54.3 | 73.1 | 72.3

31. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin ≥ 1.5% (Grouped Analysis)
Description: Clinical response at Week 26 was assessed by the percentage of participants with a decrease from Baseline in HbA1c of greater than or equal to 1.5%.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone.
Time Frame: Baseline and Week 26
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
percentage of participants | 27.6 | 45.9 | 50.3

32. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin ≥ 1.5%
Description: Clinical response at Week 26 was assessed by the percentage of participants with a decrease from Baseline in HbA1c of greater than or equal to 1.5%.
Time Frame: Baseline and Week 26
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 129 | 128 | 129 | 129 | 130 | 130 | 129 | 130 | 130 | 129 | 130 | 130
percentage of participants | 5.4 | 15.6 | 28.7 | 21.7 | 41.5 | 46.2 | 27.1 | 45.4 | 46.2 | 34.1 | 50.8 | 58.5

33. Primary Outcome: Change From Baseline to Week 26 in HbA1c
Description: The change from Baseline to Week 26 in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound).
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 126 | 122 | 123 | 127 | 130 | 127 | 123 | 128 | 124 | 126 | 127 | 126
percentage of glycosylated hemoglobin | -0.13 (0.080) | -0.64 (0.081) | -0.90 (0.081) | -0.75 (0.079) | -1.34 (0.078) | -1.27 (0.079) | -0.92 (0.081) | -1.39 (0.079) | -1.39 (0.080) | -1.00 (0.080) | -1.55 (0.079) | -1.60 (0.080)
Statistical Analysis 1: Comparison: Alogliptin 12.5 + Placebo vs Alogliptin 12.5 + Pioglitazone 15; Test type: Superiority or Other; p < 0.001, ANCOVA — As a supportive analysis, each of the individual combination treatment groups was compared with the component treatment groups receiving aloliptin alone and pioglitazone alone at the 2-sided 0.05 significance level with no multiplicity adjustment; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.70, 95% CI 2-sided [-0.93 to -0.48]
Statistical Analysis 2: Comparison: Placebo + Pioglitazone 15 vs Alogliptin 12.5 + Pioglitazone 15; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.59, 95% CI 2-sided [-0.81 to -0.38]
Statistical Analysis 3: Comparison: Alogliptin 25 + Placebo vs Alogliptin 25 + Pioglitazone 15; Test type: Superiority or Other; p = 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.37, 95% CI 2-sided [-0.59 to -0.15]
Statistical Analysis 4: Comparison: Placebo + Pioglitazone 15 vs Alogliptin 25 + Pioglitazone 15; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.52, 95% CI 2-sided [-0.74 to -0.30]
Statistical Analysis 5: Comparison: Alogliptin 12.5 + Placebo vs Alogliptin 12.5 + Pioglitazone 30; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.76, 95% CI 2-sided [-0.98 to -0.53]
Statistical Analysis 6: Comparison: Placebo + Pioglitazone 30 vs Alogliptin 12.5 + Pioglitazone 30; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.47, 95% CI 2-sided [-0.70 to -0.25]
Statistical Analysis 7: Comparison: Alogliptin 25 + Placebo vs Alogliptin 25 + Pioglitazone 30; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.49, 95% CI 2-sided [-0.71 to -0.27]
Statistical Analysis 8: Comparison: Placebo + Pioglitazone 30 vs Alogliptin 25 + Pioglitazone 30; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.47, 95% CI 2-sided [-0.70 to -0.25]
Statistical Analysis 9: Comparison: Alogliptin 12.5 + Placebo vs Alogliptin 12.5 + Pioglitazone 45; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.91, 95% CI 2-sided [-1.13 to -0.68]
Statistical Analysis 10: Comparison: Placebo + Pioglitazone 45 vs Alogliptin 12.5 + Pioglitazone 45; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.55, 95% CI 2-sided [-0.77 to -0.33]
Statistical Analysis 11: Comparison: Alogliptin 25 + Placebo vs Alogliptin 25 + Pioglitazone 45; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.70, 95% CI 2-sided [-0.92 to -0.48]
Statistical Analysis 12: Comparison: Placebo + Pioglitazone 45 vs Alogliptin 25 + Pioglitazone 45; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.61, 95% CI 2-sided [-0.83 to -0.39]

34. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin ≥ 2.0% (Grouped Analysis)
Description: Clinical response at Week 26 was assessed by the percentage of participants with a decrease from Baseline in HbA1c of greater than or equal to 2.0%.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone.
Time Frame: Baseline and Week 26.
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
percentage of participants | 11.1 | 25.4 | 27.7

35. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin ≥ 2%
Description: Clinical response at Week 26 was assessed by the percentage of participants with a decrease from Baseline in HbA1c of greater than or equal to 2%.
Time Frame: Baseline and Week 26
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 129 | 128 | 129 | 129 | 130 | 130 | 129 | 130 | 130 | 129 | 130 | 130
percentage of participants | 1.6 | 7.8 | 11.6 | 7.0 | 23.1 | 21.5 | 9.3 | 22.3 | 26.2 | 17.1 | 30.8 | 35.4

36. Secondary Outcome: Change From Baseline in Fasting Proinsulin Over Time (Grouped Analysis)
Description: Proinsulin is a precursor to insulin, and was measured as an indicator of pancreatic function. The change from Baseline in fasting proinsulin was assessed at Weeks 4, 8, 12, 16, 20 and 26.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and proinsulin as continuous covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
pmol/L
  Week 4 (n=328, 319, 327) | -6.2 (0.81) | -10.3 (0.82) | -10.1 (0.81)
  Week 8 (n=357, 347, 358) | -7.2 (0.87) | -11.3 (0.88) | -11.3 (0.87)
  Week 12 (n=357, 347, 358) | -8.2 (0.91) | -11.6 (0.93) | -11.6 (0.91)
  Week 16 (n=358, 348, 358) | -7.2 (0.92) | -12.2 (0.94) | -11.3 (0.92)
  Week 20 (n=358, 349, 359) | -6.6 (1.08) | -10.4 (1.09) | -10.7 (1.08)
  Week 26 (n=358, 349, 359) | -5.3 (1.09) | -10.6 (1.11) | -9.5 (1.09)

37. Secondary Outcome: Change From Baseline to Week 4 in Fasting Proinsulin
Description: Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline proinsulin as continuous covariates.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 116 | 111 | 109 | 107 | 109 | 109 | 110 | 105 | 114 | 111 | 105 | 104
pmol/L | -0.1 (1.36) | -4.7 (1.39) | -2.3 (1.41) | -4.8 (1.42) | -9.9 (1.41) | -8.9 (1.41) | -6.7 (1.40) | -9.6 (1.43) | -9.5 (1.37) | -7.2 (1.39) | -11.3 (1.43) | -11.7 (1.44)

38. Secondary Outcome: Change From Baseline to Week 8 in Fasting Proinsulin
Description: as for outcome 37
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 120 | 123 | 121 | 119 | 120 | 116 | 113 | 119 | 120 | 115 | 119
pmol/L | 0.7 (1.48) | 0.2 (1.50) | -2.6 (1.48) | -3.8 (1.49) | -11.1 (1.50) | -10.7 (1.50) | -8.8 (1.52) | -11.8 (1.54) | -9.4 (1.50) | -9.0 (1.50) | -11.0 (1.53) | -13.8 (1.50)

39. Secondary Outcome: Change From Baseline to Week 12 in Fasting Proinsulin
Description: as for outcome 37
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 120 | 123 | 121 | 119 | 120 | 116 | 113 | 119 | 120 | 115 | 119
pmol/L | -1.0 (1.56) | -0.7 (1.57) | -2.3 (1.56) | -5.3 (1.57) | -10.1 (1.58) | -8.8 (1.58) | -11.2 (1.60) | -12.1 (1.63) | -12.7 (1.58) | -8.1 (1.58) | -12.7 (1.61) | -13.2 (1.58)

40. Secondary Outcome: Change From Baseline to Week 16 in Fasting Proinsulin
Description: as for outcome 37
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 120 | 123 | 121 | 120 | 120 | 117 | 113 | 119 | 120 | 115 | 119
pmol/L | -3.0 (1.58) | 0.0 (1.60) | -2.3 (1.58) | -3.7 (1.59) | -11.0 (1.60) | -8.4 (1.60) | -10.0 (1.62) | -12.6 (1.65) | -11.2 (1.60) | -8.0 (1.60) | -13.0 (1.63) | -14.4 (1.60)

41. Secondary Outcome: Change From Baseline to Week 20 in Fasting Proinsulin
Description: as for outcome 37
Time Frame: Baseline and Week 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 120 | 123 | 121 | 121 | 121 | 117 | 113 | 119 | 120 | 115 | 119
pmol/L | -0.9 (1.85) | 1.5 (1.86) | -3.0 (1.84) | -3.4 (1.86) | -11.2 (1.86) | -8.7 (1.86) | -9.3 (1.89) | -10.0 (1.92) | -10.7 (1.87) | -7.1 (1.86) | -10.2 (1.90) | -12.5 (1.87)

42. Secondary Outcome: Change From Baseline to Week 26 in Fasting Proinsulin
Description: as for outcome 37
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 120 | 123 | 121 | 121 | 121 | 117 | 113 | 119 | 120 | 115 | 119
pmol/L | 1.2 (1.87) | 0.7 (1.88) | -3.3 (1.86) | -3.5 (1.88) | -10.9 (1.88) | -7.2 (1.88) | -8.4 (1.91) | -8.9 (1.95) | -8.8 (1.89) | -4.1 (1.89) | -12.1 (1.93) | -12.6 (1.89)

43. Secondary Outcome: Change From Baseline in Insulin Over Time (Grouped Analysis)
Description: The change from Baseline in fasting insulin was assessed at Weeks 4, 8, 12, 16, 20 and 26. This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline insulin as continuous covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: µIU/mL
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
µIU/mL
  Week 4 (n=325, 318, 326) | -2.29 (0.440) | -2.11 (0.445) | -2.19 (0.440)
  Week 8 (n=355, 346, 356) | -2.35 (0.535) | -2.44 (0.542) | -2.36 (0.534)
  Week 12 (n=355, 347, 356) | -2.62 (0.498) | -1.73 (0.503) | -2.62 (0.497)
  Week 16 (n=356, 348, 356) | -2.19 (0.488) | -2.60 (0.494) | -2.48 (0.488)
  Week 20 (n=356, 349, 357) | -2.35 (0.511) | -1.91 (0.516) | -2.06 (0.510)
  Week 26 (n=356, 349, 357) | -1.74 (1.212) | -2.05 (1.225) | -1.66 (1.210)

44. Secondary Outcome: Change From Baseline to Week 4 in Insulin Levels
Description: Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline insulin as continuous covariates.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: µIU/mL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 116 | 110 | 106 | 107 | 109 | 108 | 109 | 104 | 114 | 109 | 105 | 104
µIU/mL | 1.06 (0.737) | -0.33 (0.756) | 2.31 (0.771) | -1.68 (0.767) | -3.03 (0.760) | -1.86 (0.763) | -2.43 (0.760) | -1.45 (0.779) | -2.05 (0.743) | -2.76 (0.760) | -1.85 (0.774) | -2.65 (0.778)

45. Secondary Outcome: Change From Baseline to Week 8 in Insulin Levels
Description: as for outcome 44
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: µIU/mL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 119 | 123 | 121 | 119 | 119 | 116 | 112 | 118 | 118 | 115 | 119
µIU/mL | -0.46 (0.912) | 1.80 (0.923) | 1.69 (0.909) | -1.47 (0.916) | -2.21 (0.923) | -2.78 (0.923) | -2.74 (0.935) | -3.15 (0.953) | -1.20 (0.927) | -2.83 (0.927) | -1.96 (0.939) | -3.09 (0.924)

46. Secondary Outcome: Change From Baseline to Week 12 in Insulin Levels
Description: as for outcome 44
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: µIU/mL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 119 | 123 | 121 | 119 | 119 | 116 | 113 | 118 | 118 | 115 | 119
µIU/mL | 0.06 (0.849) | 1.79 (0.859) | 1.93 (0.846) | -1.29 (0.852) | -1.47 (0.859) | -2.01 (0.859) | -3.61 (0.870) | -1.36 (0.882) | -2.83 (0.863) | -2.95 (0.863) | -2.35 (0.874) | -3.01 (0.859)

47. Secondary Outcome: Change From Baseline to Week 16 in Insulin Levels
Description: as for outcome 44
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: µIU/mL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 119 | 123 | 121 | 120 | 119 | 117 | 113 | 118 | 118 | 115 | 119
µIU/mL | 0.34 (0.833) | 1.22 (0.843) | 1.83 (0.830) | -0.63 (0.836) | -2.28 (0.840) | -1.11 (0.843) | -3.46 (0.851) | -2.50 (0.866) | -2.82 (0.847) | -2.48 (0.847) | -3.00 (0.858) | -3.52 (0.844)

48. Secondary Outcome: Change From Baseline to Week 20 in Insulin Levels
Description: as for outcome 44
Time Frame: Baseline and Week 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: µIU/mL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 119 | 123 | 121 | 121 | 120 | 117 | 113 | 118 | 118 | 115 | 119
µIU/mL | 0.18 (0.873) | 2.03 (0.883) | 0.76 (0.869) | -0.66 (0.876) | -2.35 (0.876) | -0.90 (0.880) | -3.29 (0.891) | -2.20 (0.907) | -2.29 (0.887) | -3.12 (0.887) | -1.16 (0.899) | -3.01 (0.884)

49. Secondary Outcome: Change From Baseline to Week 26 in Insulin Levels
Description: as for outcome 44
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: µIU/mL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 119 | 123 | 121 | 121 | 120 | 117 | 113 | 118 | 118 | 115 | 119
µIU/mL | 6.78 (2.071) | 1.33 (2.096) | 1.43 (2.063) | -0.78 (2.078) | -3.05 (2.078) | -0.76 (2.087) | -2.56 (2.114) | -0.76 (2.152) | -1.42 (2.105) | -1.88 (2.105) | -2.33 (2.132) | -2.79 (2.096)

50. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio Over Time (Grouped Analysis)
Description: The ratio of proinsulin to insulin was calculated as proinsulin (pmol/L) / insulin (μIU/mL) at weeks 4, 8, 12, 16, 20 and 26 relative to the Baseline value.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline proinsulin/insulin ratio as continuous covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
ratio
  Week 4 (n=325, 315, 326) | -0.021 (0.0088) | -0.078 (0.0089) | -0.057 (0.0088)
  Week 8 (n=355, 344, 356) | -0.019 (0.0084) | -0.079 (0.0086) | -0.081 (0.0084)
  Week 12 (n=355, 345, 356) | -0.042 (0.0083) | -0.086 (0.0084) | -0.082 (0.0083)
  Week 16 (n=356, 346, 356) | -0.033 (0.0077) | -0.091 (0.0078) | -0.077 (0.0077)
  Week 20 (n=356, 347, 357) | -0.034 (0.0076) | -0.088 (0.0077) | -0.078 (0.0076)
  Week 26 (n=356, 347, 357) | -0.027 (0.0088) | -0.087 (0.0090) | -0.076 (0.0088)

51. Secondary Outcome: Change From Baseline to Week 4 in Proinsulin/Insulin Ratio
Description: The ratio of proinsulin to insulin was calculated as proinsulin (pmol/L) / insulin (μIU/mL).
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline proinsulin/insulin ratio as continuous covariates.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 116 | 110 | 106 | 107 | 108 | 108 | 109 | 102 | 114 | 109 | 105 | 104
ratio | -0.015 (0.0147) | -0.039 (0.0151) | -0.058 (0.0154) | -0.029 (0.0153) | -0.054 (0.0153) | -0.054 (0.0153) | -0.023 (0.0152) | -0.068 (0.0157) | -0.045 (0.0149) | -0.009 (0.0152) | -0.111 (0.0155) | -0.072 (0.0156)

52. Secondary Outcome: Change From Baseline to Week 8 in Proinsulin/Insulin Ratio
Description: as for outcome 51
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 119 | 123 | 121 | 119 | 119 | 116 | 110 | 118 | 118 | 115 | 119
ratio | 0.005 (0.0144) | -0.025 (0.0146) | -0.045 (0.0143) | -0.007 (0.0144) | -0.086 (0.0146) | -0.077 (0.0146) | -0.036 (0.0148) | -0.054 (0.0152) | -0.072 (0.0146) | -0.013 (0.0146) | -0.098 (0.0148) | -0.093 (0.0146)

53. Secondary Outcome: Change From Baseline to Week 12 in Proinsulin/Insulin Ratio
Description: as for outcome 51
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 119 | 123 | 121 | 119 | 119 | 116 | 111 | 118 | 118 | 115 | 119
ratio | -0.006 (0.0142) | -0.024 (0.0144) | -0.041 (0.0141) | -0.041 (0.0142) | -0.073 (0.0144) | -0.056 (0.0144) | -0.063 (0.0146) | -0.072 (0.0149) | -0.088 (0.0144) | -0.021 (0.0144) | -0.112 (0.0146) | -0.101 (0.0144)

54. Secondary Outcome: Change From Baseline to Week 16 in Proinsulin/Insulin Ratio
Description: as for outcome 51
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 119 | 123 | 121 | 120 | 119 | 117 | 111 | 118 | 118 | 115 | 119
ratio | -0.026 (0.0132) | -0.036 (0.0133) | -0.046 (0.0131) | -0.035 (0.0132) | -0.078 (0.0133) | -0.066 (0.0134) | -0.035 (0.0135) | -0.094 (0.0138) | -0.061 (0.0134) | -0.030 (0.0134) | -0.102 (0.0136) | -0.104 (0.0133)

55. Secondary Outcome: Change From Baseline to Week 20 in Proinsulin/Insulin Ratio
Description: as for outcome 51
Time Frame: Baseline and Week 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 119 | 123 | 121 | 121 | 120 | 117 | 111 | 118 | 118 | 115 | 119
ratio | -0.007 (0.0131) | -0.014 (0.0132) | -0.046 (0.0130) | -0.039 (0.0131) | -0.081 (0.0131) | -0.065 (0.0132) | -0.042 (0.0133) | -0.085 (0.0137) | -0.077 (0.0133) | -0.020 (0.0133) | -0.099 (0.0134) | -0.092 (0.0132)

56. Secondary Outcome: Change From Baseline to Week 26 in Proinsulin/Insulin Ratio
Description: as for outcome 51
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 119 | 123 | 121 | 121 | 120 | 117 | 111 | 118 | 118 | 115 | 119
ratio | -0.007 (0.0151) | -0.001 (0.0153) | -0.064 (0.0151) | -0.038 (0.0152) | -0.071 (0.0152) | -0.063 (0.0152) | -0.030 (0.0154) | -0.081 (0.0159) | -0.072 (0.0154) | -0.014 (0.0154) | -0.109 (0.0156) | -0.092 (0.0153)

57. Secondary Outcome: Change From Baseline in C-peptide Over Time (Grouped Analysis)
Description: C-peptide is a byproduct created when the hormone insulin is produced and is measured by a blood test. Change from Baseline was assessed at Weeks 4, 8, 12, 16, 20 and 26.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline C-peptide as continuous covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
ng/mL
  Week 4 (n=335, 335, 336) | -0.292 (0.0417) | -0.255 (0.0417) | -0.282 (0.0416)
  Week 8 (n=367, 366, 371) | -0.356 (0.0464) | -0.327 (0.0464) | -0.311 (0.0461)
  Week 12 (n=367, 369, 374) | -0.268 (0.0781) | -0.249 (0.0779) | -0.334 (0.0774)
  Week 16 (n=369, 374, 374) | -0.352 (0.0456) | -0.343 (0.0453) | -0.333 (0.0453)
  Week 20 (n=369, 375, 375) | -0.360 (0.0465) | -0.350 (0.0461) | -0.293 (0.0461)
  Week 26 (n=371, 378, 375) | -0.341 (0.0460) | -0.346 (0.0456) | -0.326 (0.0457)

58. Secondary Outcome: Change From Baseline to Week 4 in C-peptide Levels
Description: Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline C-peptide as continuous covariates.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 117 | 110 | 108 | 109 | 114 | 112 | 112 | 113 | 117 | 114 | 108 | 107
ng/mL | 0.002 (0.0705) | -0.032 (0.0727) | 0.076 (0.0734) | -0.246 (0.0730) | -0.248 (0.0714) | -0.238 (0.0720) | -0.232 (0.0721) | -0.259 (0.0718) | -0.268 (0.0705) | -0.393 (0.0714) | -0.252 (0.0734) | -0.337 (0.0738)

59. Secondary Outcome: Change From Baseline to Week 8 in C-peptide Levels
Description: as for outcome 58
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 124 | 121 | 123 | 124 | 124 | 123 | 119 | 123 | 124 | 124 | 119 | 124
ng/mL | -0.044 (0.0798) | 0.114 (0.0807) | 0.108 (0.0801) | -0.221 (0.0798) | -0.315 (0.0798) | -0.261 (0.0801) | -0.380 (0.0814) | -0.365 (0.0802) | -0.207 (0.0797) | -0.467 (0.0798) | -0.300 (0.0814) | -0.464 (0.0798)

60. Secondary Outcome: Change From Baseline to Week 12 in C-peptide Levels
Description: as for outcome 58
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 121 | 123 | 124 | 124 | 125 | 119 | 124 | 124 | 124 | 121 | 125
ng/mL | -0.055 (0.1338) | 0.083 (0.1360) | 0.140 (0.1349) | 0.116 (0.1344) | -0.155 (0.1344) | -0.215 (0.1338) | -0.439 (0.1372) | -0.212 (0.1345) | -0.326 (0.1343) | -0.483 (0.1344) | -0.381 (0.1360) | -0.464 (0.1339)

61. Secondary Outcome: Change From Baseline to Week 16 in C-peptide Levels
Description: as for outcome 58
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 121 | 123 | 124 | 126 | 125 | 121 | 125 | 124 | 124 | 123 | 125
ng/mL | -0.076 (0.0783) | 0.032 (0.0796) | 0.101 (0.0789) | -0.242 (0.0786) | -0.282 (0.0780) | -0.184 (0.0783) | -0.410 (0.0796) | -0.318 (0.0783) | -0.306 (0.0786) | -0.404 (0.0786) | -0.431 (0.0789) | -0.510 (0.0783)

62. Secondary Outcome: Change From Baseline to Week 20 in C-peptide Levels
Description: as for outcome 58
Time Frame: Baseline and Week 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 121 | 123 | 124 | 127 | 126 | 121 | 125 | 124 | 124 | 123 | 125
ng/mL | -0.046 (0.0799) | 0.114 (0.0812) | 0.019 (0.0805) | -0.193 (0.0802) | -0.377 (0.0792) | -0.184 (0.0795) | -0.380 (0.0812) | -0.343 (0.0799) | -0.266 (0.0802) | -0.506 (0.0802) | -0.329 (0.0805) | -0.430 (0.0799)

63. Secondary Outcome: Change From Baseline to Week 26 in C-peptide Levels
Description: as for outcome 58
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 122 | 123 | 125 | 128 | 126 | 121 | 126 | 124 | 125 | 124 | 125
ng/mL | -0.011 (0.0793) | 0.000 (0.0802) | 0.059 (0.0799) | -0.239 (0.0792) | -0.380 (0.0783) | -0.204 (0.0789) | -0.353 (0.0805) | -0.235 (0.0790) | -0.300 (0.0795) | -0.429 (0.0793) | -0.421 (0.0796) | -0.474 (0.0793)

64. Secondary Outcome: Change From Baseline in Total Cholesterol Over Time (Grouped Analysis)
Description: Change from Baseline in total cholesterol was assessed at Weeks 4, 8, 12, 16, 20 and 26. This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline total cholesterol as continuous covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
mg/dL
  Week 4 (n=345, 354, 348) | 1.6 (1.41) | -4.3 (1.39) | -6.5 (1.40)
  Week 8 (n=374, 380, 376) | 4.8 (1.42) | -1.8 (1.41) | -3.3 (1.42)
  Week 12 (n=374, 380, 376) | 6.6 (1.47) | 1.3 (1.46) | -1.7 (1.46)
  Week 16 (n=374, 380, 376) | 6.5 (1.52) | 1.2 (1.51) | 0.1 (1.51)
  Week 20 (n=374, 380, 376) | 5.9 (1.56) | 3.0 (1.55) | 1.5 (1.56)
  Week 26 (n=374, 380, 376) | 8.0 (1.63) | 4.4 (1.61) | 3.9 (1.62)

65. Secondary Outcome: Change From Baseline to Week 4 in Total Cholesterol Levels
Description: Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline total cholesterol as continuous covariates.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 119 | 112 | 111 | 112 | 117 | 118 | 117 | 121 | 118 | 116 | 116 | 112
mg/dL | 1.3 (2.40) | -3.8 (2.47) | -3.7 (2.48) | 2.1 (2.47) | -2.3 (2.42) | -10.2 (2.41) | 3.7 (2.42) | -7.2 (2.38) | -2.7 (2.41) | -1.2 (2.43) | -3.6 (2.43) | -6.7 (2.47)

66. Secondary Outcome: Change From Baseline to Week 8 in Total Cholesterol Levels
Description: as for outcome 65
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 121 | 123 | 125 | 128 | 127 | 123 | 127 | 124 | 126 | 125 | 125
mg/dL | 10.9 (2.46) | -1.4 (2.50) | -0.3 (2.48) | 7.3 (2.46) | -2.3 (2.43) | -4.1 (2.44) | 6.6 (2.48) | 0.1 (2.45) | 0.3 (2.47) | 0.3 (2.45) | -3.1 (2.46) | -6.2 (2.46)

67. Secondary Outcome: Change From Baseline to Week 12 in Total Cholesterol Levels
Description: as for outcome 65
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 122 | 123 | 125 | 128 | 127 | 123 | 127 | 124 | 126 | 125 | 125
mg/dL | 7.8 (2.54) | 0.4 (2.57) | 0.1 (2.56) | 8.7 (2.54) | 1.9 (2.51) | -0.2 (2.52) | 7.3 (2.56) | 0.3 (2.52) | -1.0 (2.55) | 3.7 (2.53) | 1.7 (2.54) | -3.9 (2.54)

68. Secondary Outcome: Change From Baseline to Week 16 in Total Cholesterol Levels
Description: as for outcome 65
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 122 | 123 | 125 | 128 | 127 | 123 | 127 | 124 | 126 | 125 | 125
mg/dL | 5.0 (2.62) | -0.5 (2.66) | -2.9 (2.65) | 7.2 (2.62) | -0.4 (2.59) | 3.2 (2.60) | 10.0 (2.65) | 0.9 (2.61) | -1.2 (2.63) | 2.3 (2.61) | 2.9 (2.62) | -1.8 (2.62)

69. Secondary Outcome: Change From Baseline to Week 20 in Total Cholesterol Levels
Description: as for outcome 65
Time Frame: Baseline and Week 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 122 | 123 | 125 | 128 | 127 | 123 | 127 | 124 | 126 | 125 | 125
mg/dL | 6.7 (2.70) | 1.8 (2.74) | -1.9 (2.73) | 6.3 (2.70) | 4.0 (2.67) | 1.4 (2.68) | 7.0 (2.73) | 1.1 (2.68) | 3.4 (2.71) | 4.6 (2.69) | 4.0 (2.70) | -0.3 (2.70)

70. Secondary Outcome: Change From Baseline to Week 26 in Total Cholesterol Levels
Description: as for outcome 65
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 122 | 123 | 125 | 128 | 127 | 123 | 127 | 124 | 126 | 125 | 125
mg/dL | 4.4 (2.82) | 2.2 (2.85) | 0.9 (2.84) | 5.8 (2.81) | 4.3 (2.78) | 3.5 (2.79) | 8.8 (2.84) | 2.8 (2.80) | 3.2 (2.83) | 9.5 (2.80) | 6.0 (2.81) | 5.1 (2.81)

71. Secondary Outcome: Change From Baseline in Low-Density Lipoprotein Cholesterol Over Time (Grouped Analysis)
Description: Change from Baseline in low-density lipoprotein cholesterol (LDL-C) was assessed at Weeks 4, 8, 12, 16, 20 and 26.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline LDL cholesterol as continuous covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
mg/dL
  Week 4 (n=330, 336, 338) | 3.1 (1.23) | -0.5 (1.22) | -1.9 (1.22)
  Week 8 (n=365, 365, 365) | 5.9 (1.28) | 1.3 (1.28) | 0.1 (1.28)
  Week 12 (n=365, 367, 366) | 6.9 (1.29) | 3.3 (1.29) | 1.5 (1.29)
  Week 16 (n=365, 368, 366) | 6.1 (1.29) | 3.3 (1.29) | 2.4 (1.29)
  Week 20 (n=365, 368, 366) | 6.9 (1.37) | 4.2 (1.36) | 3.0 (1.37)
  Week 26 (n=365, 368, 366) | 7.4 (1.39) | 5.2 (1.39) | 5.6 (1.39)

72. Secondary Outcome: Change From Baseline to Week 4 in Low-Density Lipoprotein Cholesterol
Description: Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline LDL cholesterol as continuous covariates.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 113 | 102 | 105 | 107 | 112 | 113 | 112 | 115 | 114 | 111 | 109 | 111
mg/dL | 2.1 (2.11) | -2.4 (2.22) | 1.4 (2.19) | 2.6 (2.16) | 1.6 (2.12) | -2.7 (2.11) | 3.2 (2.12) | -2.8 (2.09) | 0.4 (2.10) | 3.4 (2.13) | -0.3 (2.15) | -3.4 (2.13)

73. Secondary Outcome: Change From Baseline to Week 8 in Low-Density Lipoprotein Cholesterol
Description: as for outcome 72
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 119 | 113 | 119 | 122 | 123 | 122 | 120 | 123 | 119 | 123 | 119 | 124
mg/dL | 9.4 (2.24) | 2.1 (2.30) | 3.4 (2.24) | 7.3 (2.21) | -0.4 (2.21) | 1.0 (2.21) | 5.4 (2.24) | 2.4 (2.21) | 2.7 (2.24) | 4.8 (2.21) | 2.0 (2.24) | -3.2 (2.20)

74. Secondary Outcome: Change From Baseline to Week 12 in Low-Density Lipoprotein Cholesterol
Description: as for outcome 72
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 120 | 115 | 119 | 122 | 125 | 122 | 120 | 123 | 120 | 123 | 119 | 124
mg/dL | 6.5 (2.26) | 1.9 (2.30) | 3.7 (2.26) | 8.9 (2.24) | 3.3 (2.21) | 3.8 (2.24) | 6.1 (2.26) | 1.9 (2.23) | 0.9 (2.25) | 5.7 (2.23) | 4.9 (2.26) | -0.3 (2.22)

75. Secondary Outcome: Change From Baseline to Week 16 in Low-Density Lipoprotein Cholesterol
Description: as for outcome 72
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 120 | 116 | 119 | 122 | 125 | 122 | 120 | 123 | 120 | 123 | 120 | 124
mg/dL | 4.2 (2.25) | 1.3 (2.29) | 0.9 (2.26) | 7.1 (2.23) | 2.9 (2.21) | 4.6 (2.23) | 7.1 (2.25) | 2.1 (2.23) | 0.8 (2.25) | 4.1 (2.22) | 4.9 (2.25) | 1.8 (2.21)

76. Secondary Outcome: Change From Baseline to Week 20 in Low-Density Lipoprotein Cholesterol
Description: as for outcome 72
Time Frame: Baseline and Week 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 120 | 116 | 119 | 122 | 125 | 122 | 120 | 123 | 120 | 123 | 120 | 124
mg/dL | 6.9 (2.39) | 2.9 (2.43) | 1.9 (2.40) | 7.7 (2.37) | 4.3 (2.34) | 3.0 (2.37) | 6.6 (2.39) | 2.3 (2.36) | 4.1 (2.39) | 6.3 (2.36) | 6.1 (2.39) | 1.9 (2.35)

77. Secondary Outcome: Change From Baseline to Week 26 in Low-Density Lipoprotein Cholesterol
Description: as for outcome 72
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 120 | 116 | 119 | 122 | 125 | 122 | 120 | 123 | 120 | 123 | 120 | 124
mg/dL | 3.6 (2.43) | 2.8 (2.47) | 3.6 (2.44) | 7.9 (2.41) | 3.7 (2.38) | 6.1 (2.41) | 6.2 (2.43) | 2.9 (2.40) | 3.0 (2.43) | 8.1 (2.40) | 9.1 (2.43) | 7.7 (2.39)

78. Secondary Outcome: Change From Baseline in High-Density Lipoprotein Cholesterol Over Time (Grouped Analysis)
Description: Change from Baseline in high-density lipoprotein cholesterol (HDL-C) was assessed at Weeks 4, 8, 12, 16, 20 and 26.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline HDL cholesterol as continuous covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
mg/dL
  Week 4 (n=345, 353, 348) | 3.0 (0.33) | 2.7 (0.33) | 3.4 (0.33)
  Week 8 (n=374, 380, 376) | 4.0 (0.35) | 4.1 (0.34) | 4.6 (0.35)
  Week 12 (n=374, 380, 376) | 5.4 (0.37) | 5.3 (0.37) | 5.1 (0.37)
  Week 16 (n=374, 380, 376) | 5.2 (0.39) | 5.2 (0.38) | 5.0 (0.38)
  Week 20 (n=374, 380, 376) | 5.2 (0.40) | 5.7 (0.40) | 5.2 (0.40)
  Week 26 (n=374, 380, 376) | 5.1 (0.41) | 5.5 (0.41) | 5.0 (0.41)

79. Secondary Outcome: Change From Baseline to Week 4 in High-Density Lipoprotein Cholesterol
Description: Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline HDL cholesterol as continuous covariates.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 119 | 112 | 111 | 112 | 116 | 118 | 117 | 121 | 118 | 116 | 116 | 112
mg/dL | -0.4 (0.57) | -0.6 (0.59) | -0.5 (0.59) | 2.5 (0.59) | 1.6 (0.58) | 1.6 (0.57) | 3.2 (0.57) | 2.3 (0.56) | 3.5 (0.57) | 3.3 (0.58) | 4.2 (0.58) | 5.1 (0.59)

80. Secondary Outcome: Change From Baseline to Week 8 in High-Density Lipoprotein Cholesterol
Description: as for outcome 79
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 121 | 123 | 125 | 128 | 127 | 123 | 127 | 124 | 126 | 125 | 125
mg/dL | -0.5 (0.60) | -0.1 (0.61) | 0.6 (0.61) | 2.8 (0.60) | 2.3 (0.59) | 2.9 (0.60) | 4.8 (0.61) | 4.2 (0.60) | 4.6 (0.60) | 4.5 (0.60) | 5.7 (0.60) | 6.3 (0.60)

81. Secondary Outcome: Change From Baseline to Week 12 in High-Density Lipoprotein Cholesterol
Description: as for outcome 79
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 122 | 123 | 125 | 128 | 127 | 123 | 127 | 124 | 126 | 125 | 125
mg/dL | -0.2 (0.64) | 0.0 (0.65) | 0.3 (0.64) | 3.8 (0.64) | 3.7 (0.63) | 3.7 (0.63) | 6.3 (0.64) | 5.8 (0.63) | 5.3 (0.64) | 6.1 (0.63) | 6.3 (0.64) | 6.4 (0.64)

82. Secondary Outcome: Change From Baseline to Week 16 in High-Density Lipoprotein Cholesterol
Description: as for outcome 79
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 122 | 123 | 125 | 128 | 127 | 123 | 127 | 124 | 126 | 125 | 125
mg/dL | -0.3 (0.67) | 0.4 (0.68) | 0.7 (0.67) | 3.9 (0.67) | 4.2 (0.66) | 4.0 (0.66) | 5.7 (0.67) | 5.5 (0.66) | 4.3 (0.67) | 5.9 (0.66) | 6.1 (0.67) | 6.7 (0.67)

83. Secondary Outcome: Change From Baseline to Week 20 in High-Density Lipoprotein Cholesterol
Description: as for outcome 79
Time Frame: Baseline and Week 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 122 | 123 | 125 | 128 | 127 | 123 | 127 | 124 | 126 | 125 | 125
mg/dL | 0.6 (0.70) | 0.9 (0.71) | 0.5 (0.70) | 3.8 (0.70) | 4.3 (0.69) | 3.9 (0.69) | 5.9 (0.70) | 5.7 (0.69) | 5.3 (0.70) | 5.9 (0.70) | 7.1 (0.70) | 6.5 (0.70)

84. Secondary Outcome: Change From Baseline to Week 26 in High-Density Lipoprotein Cholesterol
Description: as for outcome 79
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 122 | 123 | 125 | 128 | 127 | 123 | 127 | 124 | 126 | 125 | 125
mg/dL | 0.5 (0.71) | 0.6 (0.72) | 1.3 (0.71) | 3.8 (0.71) | 4.2 (0.70) | 4.1 (0.70) | 5.5 (0.71) | 6.0 (0.70) | 5.0 (0.71) | 6.1 (0.70) | 6.2 (0.71) | 6.0 (0.71)

85. Secondary Outcome: Change From Baseline in Triglycerides Over Time (Grouped Analysis)
Description: Change from Baseline in triglycerides was assessed at Weeks 4, 8, 12, 16, 20 and 26. This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline triglycerides as continuous covariates.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
mg/dL
  Week 4 (n=345, 354, 348) | -31.5 (4.07) | -38.9 (4.02) | -48.0 (4.06)
  Week 8 (n=374, 380, 376) | -34.7 (4.37) | -44.4 (4.34) | -47.9 (4.36)
  Week 12 (n=374, 380, 376) | -34.5 (4.25) | -47.5 (4.21) | -49.4 (4.24)
  Week 16 (n=374, 380, 376) | -29.4 (4.43) | -49.3 (4.39) | -46.3 (4.42)
  Week 20 (n=374, 380, 376) | -34.9 (4.30) | -43.6 (4.27) | -42.7 (4.29)
  Week 26 (n=374, 380, 376) | -29.6 (4.42) | -41.4 (4.39) | -40.7 (4.41)

86. Secondary Outcome: Change From Baseline to Week 4 in Triglyceride Levels
Description: Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline triglycerides as continuous covariates.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 119 | 112 | 111 | 112 | 117 | 118 | 117 | 121 | 118 | 116 | 116 | 112
mg/dL | -2.4 (6.93) | -2.2 (7.15) | -25.0 (7.18) | -21.5 (7.14) | -35.8 (6.99) | -51.1 (6.96) | -26.7 (6.99) | -42.2 (6.88) | -44.4 (6.96) | -47.1 (7.02) | -39.2 (7.03) | -49.1 (7.15)

87. Secondary Outcome: Change From Baseline to Week 8 in Triglyceride Levels
Description: as for outcome 86
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 121 | 123 | 125 | 128 | 127 | 123 | 127 | 124 | 126 | 125 | 125
mg/dL | 26.3 (7.56) | -16.4 (7.69) | -23.0 (7.62) | -20.5 (7.56) | -30.1 (7.47) | -46.4 (7.50) | -30.3 (7.62) | -43.1 (7.51) | -44.5 (7.60) | -53.1 (7.53) | -60.1 (7.57) | -52.7 (7.56)

88. Secondary Outcome: Change From Baseline to Week 12 in Triglyceride Levels
Description: as for outcome 86
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 122 | 123 | 125 | 128 | 127 | 123 | 127 | 124 | 126 | 125 | 125
mg/dL | 18.9 (7.35) | -4.3 (7.44) | -18.1 (7.41) | -24.1 (7.34) | -37.4 (7.26) | -44.0 (7.29) | -37.4 (7.40) | -47.9 (7.29) | -46.8 (7.38) | -42.1 (7.31) | -57.1 (7.35) | -57.4 (7.35)

89. Secondary Outcome: Change From Baseline to Week 16 in Triglyceride Levels
Description: as for outcome 86
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 122 | 123 | 125 | 128 | 127 | 123 | 127 | 124 | 126 | 125 | 125
mg/dL | 10.6 (7.66) | -7.5 (7.75) | -26.8 (7.72) | -10.5 (7.66) | -53.0 (7.57) | -33.8 (7.60) | -28.2 (7.72) | -44.2 (7.60) | -45.9 (7.69) | -49.4 (7.63) | -50.7 (7.66) | -59.1 (7.66)

90. Secondary Outcome: Change From Baseline to Week 20 in Triglyceride Levels
Description: as for outcome 86
Time Frame: Baseline and Week 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 122 | 123 | 125 | 128 | 127 | 123 | 127 | 124 | 126 | 125 | 125
mg/dL | 5.7 (7.44) | -7.0 (7.53) | -23.7 (7.50) | -18.0 (7.44) | -41.2 (7.35) | -34.6 (7.38) | -37.5 (7.50) | -43.1 (7.39) | -42.4 (7.47) | -49.3 (7.41) | -46.4 (7.44) | -51.2 (7.44)

91. Secondary Outcome: Change From Baseline to Week 26 in Triglyceride Levels
Description: as for outcome 86
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 125 | 122 | 123 | 125 | 128 | 127 | 123 | 127 | 124 | 126 | 125 | 125
mg/dL | 3.7 (7.65) | -1.1 (7.74) | -15.2 (7.71) | -29.5 (7.65) | -37.7 (7.56) | -38.5 (7.59) | -27.0 (7.71) | -37.3 (7.59) | -33.5 (7.68) | -32.4 (7.62) | -49.3 (7.65) | -50.1 (7.65)

92. Secondary Outcome: Change From Baseline in Free Fatty Acids Over Time (Grouped Analysis)
Description: Change from Baseline in free fatty acids (FFA) was assessed at Weeks 12 and 26. This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline free fatty acid as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
mmol/L
  Week 12 (n=339, 356, 352) | -0.0707 (0.01483) | -0.1306 (0.01447) | -0.1273 (0.01455)
  Week 26 (n=353, 368, 363) | -0.0676 (0.01050) | -0.0945 (0.01029) | -0.1144 (0.01036)

93. Secondary Outcome: Change From Baseline to Week 12 in Free Fatty Acids
Description: Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline free fatty acid as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 120 | 116 | 116 | 115 | 119 | 118 | 111 | 118 | 116 | 113 | 119 | 118
mmol/L | 0.0067 (0.02493) | -0.0149 (0.02535) | -0.0769 (0.02535) | -0.0879 (0.02547) | -0.1305 (0.02502) | -0.1291 (0.02512) | -0.0395 (0.02592) | -0.1167 (0.02515) | -0.1126 (0.02534) | -0.0848 (0.02567) | -0.1447 (0.02503) | -0.1401 (0.02514)

94. Secondary Outcome: Change From Baseline to Week 26 in Free Fatty Acids
Description: as for outcome 93
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 120 | 122 | 117 | 124 | 121 | 118 | 122 | 120 | 118 | 122 | 122
mmol/L | -0.0387 (0.01788) | -0.0427 (0.01802) | -0.0386 (0.01787) | -0.0561 (0.01825) | -0.0752 (0.01772) | -0.0972 (0.01793) | -0.0737 (0.01817) | -0.0956 (0.01788) | -0.1232 (0.01801) | -0.0730 (0.01816) | -0.1125 (0.01787) | -0.1228 (0.01787)

95. Secondary Outcome: Change From Baseline in Plasminogen Activator Inhibitor-1 Over Time (Grouped Analysis)
Description: Change from Baseline in plasminogen activator inhibitor-1 (PAI-1) was assessed at Weeks 12 and 26.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline PAI-1 as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
ng/mL
  Week 12 (n=311, 333, 328) | -4.14 (1.970) | -8.76 (1.900) | -8.57 (1.914)
  Week 26 (n=341, 354, 348) | -4.56 (2.049) | -2.69 (2.010) | -9.25 (2.027)

96. Secondary Outcome: Change From Baseline to Week 12 in Plasminogen Activator Inhibitor-1
Description: Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline PAI-1 as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 106 | 107 | 107 | 108 | 113 | 109 | 107 | 108 | 109 | 96 | 112 | 110
ng/mL | -4.55 (3.367) | 3.54 (3.350) | -1.80 (3.353) | -5.32 (3.340) | -6.28 (3.260) | -10.94 (3.320) | -8.53 (3.353) | -10.47 (3.336) | -1.71 (3.321) | 1.85 (3.539) | -9.13 (3.277) | -12.63 (3.306)

97. Secondary Outcome: Change From Baseline to Week 26 in Plasminogen Activator Inhibitor-1
Description: as for outcome 96
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 115 | 114 | 118 | 115 | 119 | 116 | 117 | 116 | 115 | 109 | 119 | 117
ng/mL | -3.00 (3.526) | 0.57 (3.540) | -3.29 (3.481) | -5.43 (3.529) | -4.75 (3.465) | -9.62 (3.510) | -5.24 (3.495) | 1.89 (3.511) | -6.66 (3.525) | -3.02 (3.622) | -5.22 (3.466) | -11.48 (3.496)

98. Secondary Outcome: Change From Baseline in High-sensitivity C-Reactive Protein Over Time (Grouped Analysis)
Description: Change from Baseline in high-sensitivity C-Reactive Protein (hsCRP) was assessed at Weeks 12 and 26.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline hsCRP as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
mg/L
  Week 12 (n=346, 356, 355) | -2.0274 (0.32717) | -2.4653 (0.32225) | -1.9208 (0.32253)
  Week 26 (n=359, 369, 363) | -0.8889 (0.46384) | -1.7716 (0.45715) | -0.9977 (0.46059)

99. Secondary Outcome: Change From Baseline to Week 12 in High-sensitivity C-Reactive Protein
Description: Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline hsCRP as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 120 | 114 | 118 | 114 | 119 | 118 | 118 | 119 | 116 | 114 | 118 | 121
mg/L | -1.1053 (0.55528) | -1.0730 (0.56942) | 0.3516 (0.55954) | -0.9166 (0.56902) | -2.2362 (0.55706) | -2.4217 (0.55929) | -2.7023 (0.55971) | -2.2143 (0.55757) | -1.0006 (0.56412) | -2.4212 (0.57137) | -2.9032 (0.55979) | -2.2978 (0.55243)

100. Secondary Outcome: Change From Baseline to Week 26 in High-sensitivity C-Reactive Protein
Description: as for outcome 99
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 121 | 120 | 122 | 119 | 124 | 122 | 121 | 123 | 119 | 119 | 122 | 122
mg/L | -0.0550 (0.79868) | -0.6606 (0.80145) | 0.2618 (0.79488) | 0.2375 (0.80439) | -1.2490 (0.78817) | -0.9438 (0.79442) | -1.0480 (0.79805) | -1.1725 (0.79206) | 0.1697 (0.80434) | -1.8562 (0.80771) | -2.8933 (0.79515) | -2.2191 (0.79450)

101. Secondary Outcome: Change From Baseline in Adiponectin Over Time (Grouped Analysis)
Description: Change from Baseline in adiponectin was assessed at Weeks 12 and 26. This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline adiponectin as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: μg/mL
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
μg/mL
  Week 12 (n=339, 357, 348) | 6.03 (0.353) | 6.51 (0.344) | 6.51 (0.348)
  Week 26 (n=356, 369, 361) | 5.98 (0.396) | 6.43 (0.388) | 6.46 (0.393)

102. Secondary Outcome: Change From Baseline to Week 12 in Adiponectin
Description: Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline adiponectin as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: μg/mL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 120 | 114 | 115 | 116 | 121 | 117 | 111 | 118 | 114 | 112 | 118 | 117
μg/mL | 0.02 (0.593) | 0.44 (0.609) | 0.22 (0.606) | 3.54 (0.604) | 3.78 (0.591) | 2.91 (0.601) | 6.07 (0.617) | 6.31 (0.599) | 7.13 (0.609) | 8.47 (0.614) | 9.42 (0.598) | 9.46 (0.601)

103. Secondary Outcome: Change From Baseline to Week 26 in Adiponectin
Description: as for outcome 102
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: μg/mL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 120 | 121 | 119 | 126 | 121 | 118 | 122 | 119 | 119 | 121 | 121
μg/mL | 0.43 (0.676) | 0.48 (0.681) | 0.26 (0.678) | 3.30 (0.685) | 4.80 (0.664) | 2.93 (0.678) | 5.90 (0.687) | 6.30 (0.676) | 6.87 (0.684) | 8.75 (0.684) | 8.18 (0.678) | 9.59 (0.678)

104. Secondary Outcome: Change From Baseline in Body Weight Over Time (Grouped Analysis)
Description: Change from Baseline in body weight was assessed at Weeks 8, 12, 20 and 26. This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline weight as continuous covariates.
Time Frame: Baseline and Weeks 8, 12, 20 and 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
kg
  Week 8 (n=361, 372, 367) | 0.45 (0.103) | 0.34 (0.101) | 0.63 (0.102)
  Week 12 (n=368, 374, 373) | 0.56 (0.125) | 0.57 (0.124) | 0.82 (0.124)
  Week 20 (n=368, 374, 373) | 1.21 (0.152) | 1.45 (0.151) | 1.46 (0.151)
  Week 26 (n=368, 374, 373) | 1.49 (0.168) | 1.81 (0.167) | 1.87 (0.167)

105. Secondary Outcome: Change From Baseline to Week 8 in Body Weight
Description: Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline weight as continuous covariates.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 123 | 119 | 120 | 121 | 126 | 122 | 121 | 125 | 121 | 119 | 121 | 124
kg | -0.13 (0.176) | -0.05 (0.179) | -0.45 (0.178) | 0.32 (0.177) | 0.09 (0.174) | 0.22 (0.176) | 0.57 (0.177) | 0.49 (0.174) | 0.74 (0.177) | 0.46 (0.179) | 0.43 (0.177) | 0.93 (0.175)

106. Secondary Outcome: Change From Baseline to Week 12 in Body Weight
Description: as for outcome 105
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 123 | 122 | 123 | 122 | 127 | 124 | 122 | 125 | 123 | 124 | 122 | 126
kg | -0.46 (0.216) | -0.14 (0.217) | -0.56 (0.216) | 0.39 (0.217) | 0.22 (0.213) | 0.39 (0.215) | 0.75 (0.217) | 0.60 (0.215) | 0.98 (0.216) | 0.55 (0.216) | 0.88 (0.217) | 1.08 (0.214)

107. Secondary Outcome: Change From Baseline to Week 20 in Body Weight
Description: as for outcome 105
Time Frame: Baseline and Week 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 123 | 122 | 123 | 122 | 127 | 124 | 122 | 125 | 123 | 124 | 122 | 126
kg | -0.55 (0.263) | -0.08 (0.264) | -0.48 (0.263) | 0.76 (0.264) | 0.96 (0.259) | 0.85 (0.262) | 1.51 (0.264) | 1.45 (0.261) | 1.76 (0.263) | 1.35 (0.262) | 1.93 (0.264) | 1.76 (0.260)

108. Secondary Outcome: Change From Baseline to Week 26 in Body Weight
Description: as for outcome 105
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 123 | 122 | 123 | 122 | 127 | 124 | 122 | 125 | 123 | 124 | 122 | 126
kg | -0.66 (0.291) | -0.02 (0.292) | -0.67 (0.291) | 0.94 (0.292) | 1.25 (0.287) | 1.27 (0.290) | 1.88 (0.292) | 1.89 (0.289) | 2.10 (0.291) | 1.65 (0.290) | 2.30 (0.292) | 2.25 (0.288)

109. Secondary Outcome: Change From Baseline in Calculated Homeostatic Model Assessment Insulin Resistance (HOMA IR) (Grouped Analysis)
Description: HOMA IR measures insulin resistance based on fasting glucose and insulin measurements:
  HOMA IR = fasting plasma insulin (µIU/mL) * fasting plasma glucose (mmol/L) / 22.5.
  A higher number indicates a greater insulin resistance. This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone.
  Least Squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and HOMA-IR as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: insulin resistance
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
insulin resistance
  Week 12 (n=347, 344, 351) | -1.832 (0.3122) | -1.966 (0.3136) | -2.572 (0.3104)
  Week 26 (n=348, 346, 352) | -1.571 (0.3501) | -2.209 (0.3512) | -1.711 (0.3481)

110. Secondary Outcome: Change From Baseline to Week 12 in Calculated HOMA Insulin Resistance
Description: The Homeostasis Model Assessment of insulin resistance (HOMA IR) measures insulin resistance based on fasting glucose and insulin measurements:
  HOMA IR = fasting plasma insulin (µIU/mL) * fasting plasma glucose (mmol/L) / 22.5.
  A higher number indicates a greater degree of insulin resistance. Least Squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and HOMA-IR as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: insulin resistance
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 119 | 117 | 122 | 119 | 117 | 118 | 114 | 113 | 116 | 114 | 114 | 117
insulin resistance | 0.337 (0.5333) | 0.063 (0.5375) | 0.041 (0.5270) | -1.012 (0.5330) | -1.819 (0.5376) | -2.305 (0.5352) | -2.278 (0.5446) | -1.457 (0.5473) | -2.665 (0.5400) | -2.202 (0.5447) | -2.615 (0.5446) | -2.742 (0.5377)

111. Secondary Outcome: Change From Baseline to Week 26 in Calculated HOMA Insulin Resistance
Description: as for outcome 110
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: insulin resistance
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 119 | 117 | 122 | 119 | 119 | 119 | 115 | 113 | 116 | 114 | 114 | 117
insulin resistance | 0.464 (0.5988) | 0.311 (0.6036) | -0.179 (0.5918) | -0.864 (0.5985) | -2.300 (0.5986) | -0.223 (0.5985) | -2.061 (0.6089) | -1.871 (0.6147) | -2.056 (0.6064) | -1.789 (0.6117) | -2.456 (0.6116) | -2.854 (0.6038)

112. Secondary Outcome: Change From Baseline in Homeostatic Model Assessment Beta Cell Function (Grouped Analysis)
Description: The homeostatic model assessment estimates steady state beta cell function as a percentage of a normal reference population (%B).
  HOMA %B = 20 * insulin (µIU/mL) / fasting plasma glucose (mmol/L) - 3.5.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline HOMA beta cell function as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage beta cell function
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
percentage beta cell function
  Week 12 (n=347, 344, 350) | 2.591 (3.7892) | 23.799 (3.8017) | 19.477 (3.7685)
  Week 26 (n=348, 346, 351) | 5.060 (3.0460) | 18.173 (3.0522) | 22.182 (3.0297)

113. Secondary Outcome: Change From Baseline to Week 12 in Calculated HOMA Beta-cell Function
Description: The Homeostasis Model Assessment (HOMA) estimates steady state beta cell function (%B) as a percentage of a normal reference population.
  HOMA %B = 20 * insulin (µIU/mL) / fasting plasma glucose (mmol/L) - 3.5. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline HOMA beta cell function as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage beta cell function
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 118 | 117 | 122 | 119 | 117 | 118 | 114 | 113 | 116 | 114 | 114 | 116
percentage beta cell function | -3.027 (6.4915) | 16.304 (6.5165) | 22.996 (6.3854) | 2.565 (6.4614) | 30.346 (6.5157) | 19.887 (6.4916) | 1.118 (6.6030) | 21.045 (6.6358) | 19.935 (6.5444) | 4.023 (6.6240) | 19.938 (6.6025) | 18.541 (6.5456)

114. Secondary Outcome: Change From Baseline to Week 26 in Calculated HOMA Beta-cell Function
Description: as for outcome 113
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage beta cell function
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 118 | 117 | 122 | 119 | 119 | 119 | 115 | 113 | 116 | 114 | 114 | 116
percentage beta cell function | -0.924 (5.2260) | 11.812 (5.2462) | 17.814 (5.1407) | 2.770 (5.2018) | 10.977 (5.2010) | 19.320 (5.2044) | 8.983 (5.2921) | 22.474 (5.3423) | 23.475 (5.2687) | 3.427 (5.3327) | 21.068 (5.3154) | 23.752 (5.2696)

115. Secondary Outcome: Change From Baseline in Apolipoprotein A1 Over Time (Grouped Analysis)
Description: Change from Baseline in Apolipoprotein A1 was assessed at Weeks 12 and 26. This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline apolipoprotein A1 as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
mg/dL
  Week 12 (n=339, 354, 346) | 1.4 (1.00) | 0.2 (0.98) | 0.3 (0.99)
  Week 26 (n=354, 367, 356) | -1.6 (1.09) | -1.5 (1.08) | -2.8 (1.09)

116. Secondary Outcome: Change From Baseline to Week 12 in Apolipoprotein A1
Description: Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline apolipoprotein A1 as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 117 | 114 | 112 | 113 | 119 | 114 | 114 | 119 | 118 | 112 | 116 | 114
mg/dL | -1.9 (1.70) | -4.4 (1.73) | -3.0 (1.74) | 0.8 (1.73) | -1.3 (1.69) | 1.7 (1.72) | 3.5 (1.72) | 0.7 (1.69) | 0.4 (1.69) | -0.1 (1.74) | 1.1 (1.71) | -1.2 (1.72)

117. Secondary Outcome: Change From Baseline to Week 26 in Apolipoprotein A1
Description: as for outcome 116
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 120 | 118 | 119 | 117 | 125 | 116 | 119 | 122 | 121 | 118 | 120 | 119
mg/dL | -4.9 (1.88) | -3.0 (1.90) | -4.2 (1.89) | -3.3 (1.90) | -3.5 (1.84) | -2.9 (1.91) | -0.2 (1.89) | -0.1 (1.86) | -3.2 (1.87) | -1.4 (1.89) | -1.0 (1.88) | -2.2 (1.89)

118. Secondary Outcome: Change From Baseline in Apolipoprotein A2 Over Time (Grouped Analysis)
Description: Change from Baseline in Apolipoprotein A2 was assessed at Weeks 12 and 26. This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline apolipoprotein A2 as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
mg/dL
  Week 12 (n=339, 354, 345) | 3.1 (0.26) | 2.5 (0.26) | 2.3 (0.26)
  Week 26 (n=354, 367, 355) | 2.4 (0.28) | 2.1 (0.27) | 1.8 (0.28)

119. Secondary Outcome: Change From Baseline to Week 12 in Apolipoprotein A2
Description: Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline apolipoprotein A2 as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 117 | 114 | 112 | 113 | 119 | 114 | 114 | 119 | 117 | 112 | 116 | 114
mg/dL | 0.4 (0.44) | 0.1 (0.45) | 0.4 (0.45) | 2.4 (0.45) | 1.4 (0.44) | 1.9 (0.45) | 3.7 (0.45) | 2.5 (0.44) | 1.8 (0.44) | 3.0 (0.45) | 3.7 (0.45) | 3.2 (0.45)

120. Secondary Outcome: Change From Baseline to Week 26 in Apolipoprotein A2
Description: as for outcome 119
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 120 | 118 | 119 | 117 | 125 | 116 | 119 | 122 | 120 | 118 | 120 | 119
mg/dL | 0.1 (0.47) | 0.2 (0.48) | 0.4 (0.48) | 1.9 (0.48) | 1.2 (0.47) | 1.0 (0.48) | 2.7 (0.48) | 2.1 (0.47) | 1.6 (0.47) | 2.8 (0.48) | 3.1 (0.47) | 2.7 (0.48)

121. Secondary Outcome: Change From Baseline in Apolipoprotein B Over Time (Grouped Analysis)
Description: Change from Baseline in Apolipoprotein B was assessed at Weeks 12 and 26. This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline apolipoprotein B as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
mg/dL
  Week 12 (n=338, 354, 346) | -3.0 (1.09) | -7.9 (1.06) | -10.0 (1.07)
  Week 26 (n=354, 367, 356) | -2.8 (1.16) | -6.4 (1.14) | -6.4 (1.15)

122. Secondary Outcome: Change From Baseline to Week 12 in Apolipoprotein B
Description: Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline apolipoprotein B as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 117 | 114 | 112 | 113 | 119 | 114 | 114 | 119 | 118 | 111 | 116 | 114
mg/dL | 5.0 (1.85) | -2.3 (1.87) | -3.6 (1.89) | -0.3 (1.88) | -7.2 (1.83) | -6.1 (1.87) | -2.1 (1.88) | -8.4 (1.83) | -12.2 (1.84) | -6.6 (1.90) | -8.0 (1.86) | -11.7 (1.87)

123. Secondary Outcome: Change From Baseline to Week 26 in Apolipoprotein B
Description: as for outcome 122
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 120 | 118 | 119 | 117 | 125 | 116 | 119 | 122 | 121 | 118 | 120 | 119
mg/dL | 0.6 (1.99) | -0.6 (2.00) | -3.7 (2.00) | -1.5 (2.01) | -6.0 (1.95) | -4.8 (2.02) | -3.2 (2.00) | -7.2 (1.97) | -8.8 (1.98) | -3.6 (2.00) | -6.1 (1.99) | -5.5 (2.00)

124. Secondary Outcome: Change From Baseline in Apolipoprotein C-III Over Time (Grouped Analysis)
Description: Change from Baseline in apolipoprotein C-III was assessed at Weeks 12 and 26. This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline apolipoprotein C-III as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
mg/dL
  Week 12 (n=337, 352, 345) | -0.6 (0.17) | -1.2 (0.16) | -1.3 (0.17)
  Week 26 (n=353, 366, 355) | -0.1 (0.19) | -0.6 (0.19) | -0.6 (0.19)

125. Secondary Outcome: Change From Baseline to Week 12 in Apolipoprotein C-III
Description: Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline apolipoprotein C-III as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 117 | 114 | 112 | 113 | 118 | 114 | 113 | 118 | 118 | 111 | 116 | 113
mg/dL | 0.7 (0.28) | -0.4 (0.29) | -0.7 (0.29) | -0.3 (0.29) | -1.0 (0.28) | -1.4 (0.29) | -0.3 (0.29) | -1.0 (0.28) | -1.3 (0.28) | -1.1 (0.29) | -1.4 (0.29) | -1.2 (0.29)

126. Secondary Outcome: Change From Baseline to Week 26 in Apolipoprotein C-III
Description: as for outcome 125
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 120 | 118 | 119 | 117 | 125 | 116 | 119 | 121 | 121 | 117 | 120 | 118
mg/dL | 0.4 (0.33) | 0.5 (0.33) | -0.7 (0.33) | -0.4 (0.33) | -0.6 (0.32) | -0.7 (0.33) | 0.2 (0.33) | -0.4 (0.32) | -0.6 (0.32) | 0.0 (0.33) | -0.7 (0.33) | -0.5 (0.33)

127. Secondary Outcome: Change From Baseline in Nuclear Magnetic Resonance Lipid Fractionation Total Triglycerides Over Time (Grouped Analysis)
Description: Nuclear Magnetic Resonance (NMR) lipid fractionation was used to assess the change from Baseline in total triglyceride levels at Weeks 12 and 26.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline NMR total triglycerides as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
mg/dL
  Week 12 (n=332, 345, 343) | -19.6 (3.92) | -28.8 (3.85) | -31.5 (3.86)
  Week 26 (n=348, 359, 357) | -11.5 (4.30) | -25.4 (4.23) | -22.9 (4.24)

128. Secondary Outcome: Change From Baseline to Week 12 in NMR Lipid Fractionation Total Triglycerides
Description: NMR lipid fractionation was used to assess the change from Baseline in total triglyceride levels at Week 12.
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline NMR total triglycerides as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 119 | 113 | 114 | 113 | 114 | 117 | 110 | 113 | 110 | 109 | 118 | 116
mg/dL | 20.6 (6.56) | -4.9 (6.73) | -7.8 (6.70) | -12.9 (6.72) | -21.8 (6.70) | -27.2 (6.61) | -18.3 (6.82) | -29.8 (6.73) | -31.6 (6.82) | -27.9 (6.85) | -35.1 (6.59) | -36.0 (6.64)

129. Secondary Outcome: Change From Baseline to Week 26 in NMR Lipid Fractionation Total Triglycerides
Description: NMR lipid fractionation was used to assess the change from Baseline in total triglyceride levels at Week 26.
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline NMR total triglycerides as continuous covariates.
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 117 | 120 | 116 | 120 | 120 | 116 | 118 | 116 | 116 | 121 | 121
mg/dL | 12.4 (7.26) | 7.3 (7.42) | -6.8 (7.32) | -18.9 (7.44) | -20.4 (7.32) | -23.1 (7.32) | -6.9 (7.44) | -23.5 (7.38) | -19.7 (7.44) | -8.6 (7.44) | -32.1 (7.29) | -25.8 (7.29)

130. Secondary Outcome: Change From Baseline in Very Low Density Lipoprotein (VLDL) / Chylomicron Particles Over Time (Grouped Analysis)
Description: The change from Baseline in levels of total VLDL/chylomicron particles and large VLDL/chylomicron particles was assessed by NMR lipid fractionation at Weeks 12 and 26.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline NMR VLDL/chylomicron particles as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
nmol/L
  Total Particles - Week 12 (n=332, 345, 343) | -1.85 (1.803) | -6.40 (1.770) | -7.26 (1.775)
  Total Particles - Week 26 (n=348, 359, 357) | -1.05 (1.999) | -1.87 (1.970) | -1.31 (1.975)
  Large Particles - Week 12 (n=332, 345, 343) | -1.61 (0.289) | -2.20 (0.283) | -2.17 (0.284)
  Large Particles - Week 26 (n=348, 359, 357) | -1.05 (0.342) | -2.25 (0.337) | -1.98 (0.337)

131. Secondary Outcome: Change From Baseline to Week 12 in VLDL / Chylomicron Particles
Description: The change from Baseline in levels of total VLDL/chylomicron particles and large VLDL/chylomicron particles was assessed by NMR lipid fractionation.
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline NMR VLDL/chylomicron particles as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 119 | 113 | 114 | 113 | 114 | 117 | 110 | 113 | 110 | 109 | 118 | 116
nmol/L
  Total Particles | 5.82 (3.013) | -1.59 (3.092) | -5.32 (3.077) | 2.52 (3.089) | -3.46 (3.077) | -5.57 (3.037) | 0.45 (3.135) | -7.82 (3.092) | -6.54 (3.132) | -8.58 (3.147) | -7.99 (3.027) | -9.76 (3.051)
  Large Particles | 1.12 (0.482) | -0.42 (0.495) | -0.27 (0.493) | -1.20 (0.495) | -1.63 (0.493) | -1.81 (0.486) | -1.69 (0.502) | -2.19 (0.495) | -2.29 (0.501) | -1.97 (0.504) | -2.81 (0.484) | -2.45 (0.489)

132. Secondary Outcome: Change From Baseline to Week 26 in VLDL / Chylomicron Particles
Description: as for outcome 131
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 117 | 120 | 116 | 120 | 120 | 116 | 118 | 116 | 116 | 121 | 121
nmol/L
  Total Particles | 2.80 (3.379) | 0.59 (3.450) | -5.79 (3.405) | -2.99 (3.462) | -3.31 (3.405) | -5.15 (3.405) | 3.68 (3.464) | -0.59 (3.436) | -0.35 (3.463) | -3.83 (3.463) | -1.70 (3.394) | 1.56 (3.392)
  Large Particles | 1.31 (0.577) | 0.94 (0.589) | -0.14 (0.582) | -1.56 (0.592) | -1.71 (0.582) | -1.80 (0.582) | -0.90 (0.592) | -2.24 (0.587) | -1.79 (0.592) | -0.67 (0.592) | -2.80 (0.580) | -2.36 (0.580)

133. Secondary Outcome: Change From Baseline in VLDL / Chylomicron Triglycerides Over Time (Grouped Analysis)
Description: The change from Baseline in levels of VLDL/chylomicron triglycerides was assessed by NMR lipid fractionation at Weeks 12 and 26.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline NMR VLDL/chylomicron triglycerides as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
mg/dL
  Week 12 (n=332, 345, 343) | -20.4 (3.90) | -28.5 (3.83) | -30.3 (3.84)
  Week 26 (n=348, 359, 357) | -13.0 (4.28) | -25.4 (4.22) | -23.0 (4.23)

134. Secondary Outcome: Change From Baseline to Week 12 in VLDL / Chylomicron Triglycerides
Description: The change from Baseline in VLDL/chylomicron triglyceride levels was assessed by NMR lipid fractionation. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline NMR VLDL/chylomicron triglycerides as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 119 | 113 | 114 | 113 | 114 | 117 | 110 | 113 | 110 | 109 | 118 | 116
mg/dL | 19.9 (6.51) | -3.5 (6.69) | -6.4 (6.65) | -14.2 (6.68) | -21.1 (6.65) | -26.5 (6.56) | -19.1 (6.78) | -29.5 (6.69) | -30.1 (6.77) | -28.4 (6.80) | -35.5 (6.55) | -34.8 (6.60)

135. Secondary Outcome: Change From Baseline to Week 26 in VLDL / Chylomicron Triglycerides
Description: as for outcome 134
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 117 | 120 | 116 | 120 | 120 | 116 | 118 | 116 | 116 | 121 | 121
mg/dL | 11.9 (7.23) | 8.3 (7.39) | -7.0 (7.29) | -20.4 (7.41) | -20.4 (7.29) | -23.8 (7.29) | -8.2 (7.41) | -23.5 (7.35) | -18.9 (7.41) | -10.4 (7.41) | -32.3 (7.26) | -26.2 (7.26)

136. Secondary Outcome: Change From Baseline in VLDL Particles Over Time (Grouped Analysis)
Description: The change from Baseline in levels of medium VLDL particles and small VLDL particles was assessed by NMR fractionation at Weeks 12 and 26.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline NMR VLDL particles as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
nmol/L
  Medium Particles - Week 12 (n=332, 345, 343) | -4.44 (1.174) | -5.36 (1.152) | -7.30 (1.155)
  Medium Particles - Week 26 (n=348, 359, 357) | -2.28 (1.346) | -3.02 (1.326) | -4.88 (1.329)
  Small Particles - Week 12 (n=332, 345, 343) | 4.16 (1.053) | 1.33 (1.033) | 1.91 (1.035)
  Small Particles - Week 26 (n=348, 359, 357) | 2.30 (1.084) | 3.55 (1.067) | 5.22 (1.070)

137. Secondary Outcome: Change From Baseline to Week 12 in VLDL Particles
Description: The change from Baseline in levels of medium VLDL particles and small VLDL particles was assessed by NMR lipid fractionation.
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline NMR VLDL particles as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 119 | 113 | 114 | 113 | 114 | 117 | 110 | 113 | 110 | 109 | 118 | 116
nmol/L
  Medium Particles | 2.13 (1.962) | -1.13 (2.014) | -2.88 (2.003) | -2.25 (2.011) | -3.16 (2.004) | -6.51 (1.977) | -2.59 (2.041) | -6.70 (2.013) | -7.05 (2.039) | -8.64 (2.048) | -6.38 (1.971) | -8.50 (1.987)
  Small Particles | 2.76 (1.758) | 0.39 (1.804) | -2.30 (1.797) | 5.99 (1.803) | 1.16 (1.796) | 2.60 (1.772) | 4.39 (1.829) | 1.15 (1.806) | 2.51 (1.828) | 2.22 (1.839) | 1.80 (1.765) | 0.73 (1.780)

138. Secondary Outcome: Change From Baseline to Week 26 in VLDL Particles
Description: as for outcome 137
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 117 | 120 | 116 | 120 | 120 | 116 | 118 | 116 | 116 | 121 | 121
nmol/L
  Medium Particles | 1.54 (2.275) | 0.85 (2.324) | -2.94 (2.292) | -4.43 (2.331) | -1.78 (2.293) | -5.42 (2.292) | 0.28 (2.332) | -2.17 (2.313) | -4.38 (2.331) | -2.70 (2.331) | -5.09 (2.285) | -4.83 (2.284)
  Small Particles | 0.26 (1.831) | -0.87 (1.868) | -2.91 (1.846) | 2.83 (1.876) | -0.19 (1.845) | 1.90 (1.845) | 4.16 (1.877) | 4.07 (1.863) | 5.45 (1.876) | -0.08 (1.878) | 6.77 (1.837) | 8.33 (1.837)

139. Secondary Outcome: Change From Baseline in Mean VLDL Particle Size Over Time (Grouped Analysis)
Description: The change from Baseline in mean VLDL particle size was assessed by NMR lipid fractionation at Weeks 12 and 26.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline mean VLDL particle size as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
nm
  Week 12 (n=332, 344, 343) | -2.77 (0.398) | -2.98 (0.390) | -3.02 (0.391)
  Week 26 (n=348, 358, 357) | -2.49 (0.406) | -3.67 (0.400) | -3.26 (0.400)

140. Secondary Outcome: Change From Baseline to Week 12 in Mean VLDL Particle Size
Description: The change from Baseline in mean VLDL particle size was assessed by NMR lipid fractionation.
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline mean VLDL particle size as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 119 | 113 | 114 | 113 | 113 | 117 | 110 | 113 | 110 | 109 | 118 | 116
nm | 0.65 (0.664) | 0.12 (0.681) | -0.18 (0.678) | -2.81 (0.681) | -2.10 (0.681) | -2.56 (0.669) | -3.16 (0.690) | -2.88 (0.681) | -2.49 (0.690) | -2.37 (0.694) | -4.00 (0.666) | -4.03 (0.672)

141. Secondary Outcome: Change From Baseline to Week 26 in Mean VLDL Particle Size
Description: as for outcome 140
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 117 | 120 | 116 | 119 | 120 | 116 | 118 | 116 | 116 | 121 | 121
nm | 0.26 (0.685) | 0.52 (0.700) | 0.35 (0.691) | -2.99 (0.703) | -2.66 (0.694) | -2.36 (0.691) | -2.88 (0.703) | -3.69 (0.697) | -3.30 (0.702) | -1.60 (0.703) | -4.65 (0.688) | -4.12 (0.688)

142. Secondary Outcome: Change From Baseline in Intermediate Density Lipoprotein (IDL) Particles Over Time (Grouped Analysis)
Description: The change from Baseline in levels of IDL particles was assessed by NMR lipid fractionation at Weeks 12 and 26.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline NMR IDL particles as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
nmol/L
  Week 12 (n=332, 345, 343) | 0.4 (2.16) | -3.9 (2.12) | -5.7 (2.12)
  Week 26 (n=348, 359, 357) | 2.8 (2.16) | -4.2 (2.13) | -1.5 (2.13)

143. Secondary Outcome: Change From Baseline to Week 12 in IDL Particles
Description: The change from Baseline in levels of IDL particles was assessed by NMR lipid fractionation.
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline NMR IDL particles as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 119 | 113 | 114 | 113 | 114 | 117 | 110 | 113 | 110 | 109 | 118 | 116
nmol/L | 1.6 (3.60) | -11.1 (3.70) | -6.0 (3.68) | 5.1 (3.70) | -6.0 (3.68) | -2.3 (3.64) | -2.2 (3.75) | -6.3 (3.70) | -8.1 (3.75) | -1.5 (3.76) | 0.7 (3.62) | -6.5 (3.65)

144. Secondary Outcome: Change From Baseline to Week 26 in IDL Particles
Description: as for outcome 143
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 117 | 120 | 116 | 120 | 120 | 116 | 118 | 116 | 116 | 121 | 121
nmol/L | 5.1 (3.65) | -7.3 (3.73) | -3.2 (3.68) | 5.2 (3.74) | -2.4 (3.67) | 0.0 (3.68) | 3.0 (3.74) | -5.0 (3.71) | -5.5 (3.74) | 0.1 (3.74) | -5.0 (3.66) | 1.0 (3.66)

145. Secondary Outcome: Change From Baseline in Low Density Lipoprotein (LDL) Particles Over Time (Grouped Analysis)
Description: The change from Baseline in levels of total, large, medium-small, total small and very small LDL particles was assessed by NMR fractionation at Weeks 12 and 26.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline NMR LDL particles as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
nmol/L
  Total Particles - Week 12 (n=332, 345, 343) | -104.1 (17.46) | -180.5 (17.13) | -236.8 (17.18)
  Total Particles - Week 26 (n=348, 359, 357) | -78.2 (17.83) | -146.2 (17.55) | -182.9 (17.60)
  Large Particles - Week 12 (n=332, 345, 343) | 85.5 (10.02) | 111.6 (9.83) | 102.3 (9.85)
  Large Particles - Week 26 (n=348, 359, 357) | 95.8 (11.11) | 93.9 (10.93) | 106.1 (10.96)
  Medium-Small Particles - Week 12 (n=332, 345, 343) | -36.6 (4.11) | -55.3 (4.03) | -60.1 (4.04)
  Medium-Small Particles - Week 26 (n=348, 359, 357) | -34.3 (4.22) | -44.9 (4.16) | -49.6 (4.17)
  Total Small Particles - Week 12 (n=332, 345, 343) | -191.4 (20.32) | -287.5 (19.94) | -331.4 (20.00)
  Total Small Particles - Week 26 (n=348, 359, 357) | -178.1 (21.13) | -235.0 (20.81) | -285.9 (20.87)
  Very Small Particles - Week 12 (n=332, 345, 343) | -154.6 (16.53) | -232.3 (16.23) | -271.3 (16.27)
  Very Small Particles - Week 26 (n=348, 359, 357) | -143.6 (17.23) | -190.3 (16.97) | -236.2 (17.02)

146. Secondary Outcome: Change From Baseline to Week 12 in LDL Particles
Description: The change from Baseline in levels of total, large, medium-small, total small and very small LDL particles was assessed by NMR lipid fractionation.
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline NMR LDL particles as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 119 | 113 | 114 | 113 | 114 | 117 | 110 | 113 | 110 | 109 | 118 | 116
nmol/L
  Total Particles | 52.0 (29.17) | -39.1 (29.92) | -69.9 (29.80) | -48.8 (29.91) | -143.5 (29.79) | -175.6 (29.43) | -96.2 (30.37) | -195.8 (29.93) | -248.8 (30.31) | -167.0 (30.46) | -202.2 (29.27) | -285.8 (29.52)
  Large Particles | 4.7 (16.74) | 21.1 (17.16) | -8.0 (17.09) | 56.2 (17.15) | 73.8 (17.08) | 85.7 (16.86) | 83.9 (17.43) | 126.2 (17.18) | 105.7 (17.39) | 116.9 (17.48) | 135.2 (16.79) | 116.1 (16.95)
  Medium-Small Particles | 9.4 (6.87) | -7.7 (7.04) | -5.1 (7.02) | -20.3 (7.04) | -41.1 (7.01) | -48.0 (6.93) | -34.4 (7.14) | -58.2 (7.05) | -64.1 (7.14) | -55.4 (7.17) | -66.8 (6.89) | -68.2 (6.96)
  Total Small Particles | 45.1 (33.98) | -52.0 (34.83) | -56.5 (34.70) | -109.9 (34.83) | -211.0 (34.69) | -256.3 (34.26) | -184.1 (35.32) | -313.7 (34.85) | -345.4 (35.29) | -280.4 (35.46) | -337.9 (34.08) | -392.7 (34.38)
  Very Small Particles | 36.4 (27.65) | -44.1 (28.34) | -51.9 (28.23) | -89.2 (28.33) | -170.3 (28.22) | -207.6 (27.87) | -149.8 (28.74) | -255.7 (28.36) | -281.5 (28.72) | -225.0 (28.85) | -271.0 (27.73) | -325.0 (27.97)

147. Secondary Outcome: Change From Baseline to Week 26 in LDL Particles
Description: as for outcome 146
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 117 | 120 | 116 | 120 | 120 | 116 | 118 | 116 | 116 | 121 | 121
nmol/L
  Total Particles | 15.0 (30.11) | -14.5 (30.73) | -30.8 (30.36) | -46.3 (30.86) | -115.1 (30.35) | -119.4 (30.37) | -68.6 (30.90) | -158.9 (30.62) | -209.4 (30.85) | -119.7 (30.87) | -164.6 (30.22) | -219.9 (30.21)
  Large Particles | -23.8 (18.77) | -12.3 (19.14) | 15.3 (18.91) | 70.5 (19.22) | 63.2 (18.90) | 93.1 (18.90) | 79.3 (19.27) | 96.6 (19.09) | 102.7 (19.22) | 137.7 (19.23) | 121.9 (18.83) | 122.7 (18.83)
  Medium-Small Particles | 9.1 (7.14) | 0.0 (7.28) | -6.9 (7.20) | -25.8 (7.31) | -29.9 (7.19) | -36.2 (7.20) | -30.0 (7.32) | -47.4 (7.26) | -55.0 (7.31) | -47.1 (7.31) | -57.6 (7.16) | -57.8 (7.17)
  Total Small Particles | 32.4 (35.72) | 2.2 (36.44) | -42.9 (36.00) | -122.5 (36.59) | -175.1 (35.99) | -211.5 (36.01) | -154.9 (36.60) | -248.7 (36.31) | -304.9 (36.58) | -256.9 (36.58) | -281.1 (35.82) | -341.3 (35.82)
  Very Small Particles | 24.0 (29.13) | 2.5 (29.71) | -36.6 (29.36) | -96.3 (29.84) | -145.7 (29.35) | -174.5 (29.37) | -124.9 (29.85) | -201.6 (29.61) | -250.0 (29.83) | -209.6 (29.83) | -223.6 (29.22) | -283.9 (29.21)

148. Secondary Outcome: Change From Baseline in Mean LDL Particle Size Over Time (Grouped Analysis)
Description: The change from Baseline in mean LDL particle size was assessed by NMR lipid fractionation at Weeks 12 and 26.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone.
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline mean LDL particle size as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
nm
  Week 12 (n=332, 345, 343) | 0.43 (0.034) | 0.58 (0.034) | 0.61 (0.034)
  Week 26 (n=348, 359, 357) | 0.41 (0.036) | 0.47 (0.035) | 0.54 (0.036)

149. Secondary Outcome: Change From Baseline to Week 12 in Mean LDL Particle Size
Description: The change from Baseline in mean LDL particle size was assessed by NMR lipid fractionation.
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline mean LDL particle size as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 119 | 113 | 114 | 113 | 114 | 117 | 110 | 113 | 110 | 109 | 118 | 116
nm | -0.05 (0.057) | 0.13 (0.059) | 0.06 (0.059) | 0.25 (0.059) | 0.43 (0.059) | 0.49 (0.058) | 0.44 (0.060) | 0.61 (0.059) | 0.61 (0.060) | 0.58 (0.060) | 0.68 (0.058) | 0.73 (0.058)

150. Secondary Outcome: Change From Baseline to Week 26 in Mean LDL Particle Size
Description: as for outcome 149
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 117 | 120 | 116 | 120 | 120 | 116 | 118 | 116 | 116 | 121 | 121
nm | -0.06 (0.061) | -0.01 (0.062) | 0.07 (0.061) | 0.26 (0.062) | 0.38 (0.061) | 0.41 (0.061) | 0.38 (0.062) | 0.48 (0.062) | 0.57 (0.062) | 0.59 (0.062) | 0.55 (0.061) | 0.63 (0.061)

151. Secondary Outcome: Change From Baseline in High Density Lipoprotein (HDL) Particles Over Time (Grouped Analysis)
Description: The change from Baseline in levels of total, large, medium and small HDL particles was assessed by NMR fractionation at Weeks 12 and 26.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline NMR HDL particles as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: μMOL/L
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
μMOL/L
  Total Particles - Week 12 (n=332, 345, 343) | 0.86 (0.220) | 0.58 (0.216) | 0.43 (0.216)
  Total Particles - Week 26 (n=348, 359, 357) | 0.62 (0.235) | 1.18 (0.231) | 0.78 (0.232)
  Large Particles - Week 12 (n=332, 345, 343) | 0.89 (0.111) | 0.78 (0.109) | 0.89 (0.109)
  Large Particles - Week 26 (n=348, 359, 357) | 0.81 (0.123) | 0.90 (0.121) | 1.01 (0.122)
  Medium Particles - Week 12 (n=332, 345, 343) | 1.38 (0.195) | 1.16 (0.191) | 1.63 (0.191)
  Medium Particles - Week 26 (n=348, 359, 357) | 1.34 (0.195) | 1.10 (0.192) | 1.46 (0.192)
  Small Particles - Week 12 (n=332, 345, 343) | -1.35 (0.261) | -1.39 (0.256) | -2.12 (0.256)
  Small Particles - Week 26 (n=348, 359, 357) | -1.45 (0.261) | -0.85 (0.257) | -1.73 (0.258)

152. Secondary Outcome: Change From Baseline to Week 12 in HDL Particles
Description: The change from Baseline in levels of total, large, medium and small HDL particles was assessed by NMR lipid fractionation.
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline NMR HDL particles as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: μmol/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 119 | 113 | 114 | 113 | 114 | 117 | 110 | 113 | 110 | 109 | 118 | 116
μmol/L
  Total Particles | -0.08 (0.368) | -0.06 (0.377) | 0.16 (0.375) | 0.90 (0.377) | 0.37 (0.375) | 0.55 (0.370) | 1.29 (0.382) | 0.75 (0.377) | 0.15 (0.382) | 0.40 (0.384) | 0.63 (0.369) | 0.60 (0.372)
  Large Particles | -0.21 (0.185) | -0.29 (0.190) | -0.10 (0.189) | 0.53 (0.190) | 0.24 (0.189) | 0.50 (0.186) | 1.09 (0.192) | 0.95 (0.190) | 1.12 (0.192) | 1.06 (0.193) | 1.17 (0.186) | 1.06 (0.187)
  Medium Particles | 0.17 (0.325) | -0.24 (0.333) | -0.01 (0.332) | 0.81 (0.334) | 1.15 (0.332) | 0.65 (0.328) | 1.21 (0.338) | 0.97 (0.334) | 1.89 (0.338) | 2.06 (0.339) | 1.30 (0.326) | 2.31 (0.329)
  Small Particles | -0.07 (0.435) | 0.43 (0.447) | 0.27 (0.445) | -0.25 (0.446) | -1.09 (0.445) | -0.63 (0.439) | -0.92 (0.453) | -1.18 (0.447) | -2.82 (0.452) | -2.82 (0.455) | -1.84 (0.437) | -2.84 (0.441)

153. Secondary Outcome: Change From Baseline to Week 26 in HDL Particles
Description: as for outcome 152
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: μmol/L
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 117 | 120 | 116 | 120 | 120 | 116 | 118 | 116 | 116 | 121 | 121
μmol/L
  Total Particles | 0.18 (0.397) | 0.43 (0.405) | 1.03 (0.400) | 0.37 (0.407) | 0.77 (0.400) | 1.31 (0.400) | 0.67 (0.407) | 1.15 (0.403) | 0.26 (0.406) | 0.83 (0.407) | 1.61 (0.398) | 0.77 (0.398)
  Large Particles | 0.02 (0.208) | -0.16 (0.212) | 0.39 (0.210) | 0.53 (0.213) | 0.55 (0.210) | 0.75 (0.210) | 0.64 (0.213) | 1.13 (0.212) | 1.34 (0.213) | 1.26 (0.213) | 1.02 (0.209) | 0.95 (0.209)
  Medium Particles | 0.13 (0.330) | 0.16 (0.336) | 0.54 (0.332) | 0.81 (0.338) | 0.86 (0.332) | 0.67 (0.332) | 1.48 (0.338) | 1.47 (0.335) | 1.69 (0.337) | 1.71 (0.337) | 0.96 (0.331) | 2.01 (0.330)
  Small Particles | 0.00 (0.441) | 0.41 (0.450) | 0.10 (0.444) | -0.78 (0.452) | -0.68 (0.444) | -0.17 (0.444) | -1.35 (0.452) | -1.47 (0.448) | -2.77 (0.452) | -2.21 (0.452) | -0.40 (0.443) | -2.24 (0.442)

154. Secondary Outcome: Change From Baseline in Mean HDL Particle Size Over Time (Grouped Analysis)
Description: The change from Baseline in mean HDL particle size was assessed by NMR lipid fractionation at Weeks 12 and 26.
  This analysis compared the groupings of participants who received the combination of pioglitazone with each dose of alogliptin with the grouping of participants who received pioglitazone alone. Least squares means are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline mean HDL particle size as continuous covariates.
Time Frame: Baseline and Weeks 12 and 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Pioglitazone Alone | Alogliptin 12.5 + Pioglitazone | Alogliptin 25 + Pioglitazone
Number analyzed (Participants) | 387 | 390 | 390
nm
  Week 12 (n=332, 345, 343) | 0.11 (0.013) | 0.13 (0.013) | 0.16 (0.013)
  Week 26 (n=348, 359, 357) | 0.11 (0.015) | 0.12 (0.014) | 0.17 (0.014)

155. Secondary Outcome: Change From Baseline to Week 12 in Mean HDL Particle Size
Description: The change from Baseline in mean HDL particle size was assessed by NMR lipid fractionation. Least squares means are from are from an ANCOVA model with treatment and geographic region as class variables, and baseline metformin dose and baseline mean HDL particle size as continuous covariates.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 119 | 113 | 114 | 113 | 114 | 117 | 110 | 113 | 110 | 109 | 118 | 116
nm | 0.00 (0.023) | 0.00 (0.023) | 0.00 (0.023) | 0.06 (0.023) | 0.07 (0.023) | 0.09 (0.023) | 0.10 (0.023) | 0.15 (0.023) | 0.17 (0.023) | 0.18 (0.024) | 0.17 (0.023) | 0.21 (0.023)

156. Secondary Outcome: Change From Baseline to Week 26 in Mean HDL Particle Size
Description: as for outcome 155
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Number analyzed (Participants) | 122 | 117 | 120 | 116 | 120 | 120 | 116 | 118 | 116 | 116 | 121 | 121
nm | 0.03 (0.025) | 0.00 (0.025) | 0.07 (0.025) | 0.06 (0.025) | 0.06 (0.025) | 0.11 (0.025) | 0.10 (0.025) | 0.15 (0.025) | 0.20 (0.025) | 0.19 (0.025) | 0.16 (0.025) | 0.19 (0.025)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent until the end of the study, and from spontaneous reporting for 30 days after the end of treatment.
Description: At each study visit, the investigator assessed whether any events had occurred. Patients could report events at any other time during the study. All events, whether reported by the patient or observed by the investigator, were documented, whether or not the investigator concluded the event to be related to the drug treatment.
Arm/Group | Placebo | Alogliptin 12.5 + Placebo | Alogliptin 25 + Placebo | Placebo + Pioglitazone 15 | Alogliptin 12.5 + Pioglitazone 15 | Alogliptin 25 + Pioglitazone 15 | Placebo + Pioglitazone 30 | Alogliptin 12.5 + Pioglitazone 30 | Alogliptin 25 + Pioglitazone 30 | Placebo + Pioglitazone 45 | Alogliptin 12.5 + Pioglitazone 45 | Alogliptin 25 + Pioglitazone 45
Serious Adverse Events (participants affected / at risk) | 2/129 | 5/128 | 6/129 | 1/129 | 2/130 | 1/130 | 2/129 | 3/130 | 6/130 | 10/129 | 2/130 | 5/130
Other Adverse Events (participants affected / at risk) | 41/129 | 40/128 | 46/129 | 51/129 | 45/130 | 44/130 | 40/129 | 35/130 | 51/130 | 40/129 | 47/130 | 41/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=129) | Alogliptin 12.5 + Placebo (N=128) | Alogliptin 25 + Placebo (N=129) | Placebo + Pioglitazone 15 (N=129) | Alogliptin 12.5 + Pioglitazone 15 (N=130) | Alogliptin 25 + Pioglitazone 15 (N=130) | Placebo + Pioglitazone 30 (N=129) | Alogliptin 12.5 + Pioglitazone 30 (N=130) | Alogliptin 25 + Pioglitazone 30 (N=130) | Placebo + Pioglitazone 45 (N=129) | Alogliptin 12.5 + Pioglitazone 45 (N=130) | Alogliptin 25 + Pioglitazone 45 (N=130)
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Migraine with aura (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung cyst benign (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=129) | Alogliptin 12.5 + Placebo (N=128) | Alogliptin 25 + Placebo (N=129) | Placebo + Pioglitazone 15 (N=129) | Alogliptin 12.5 + Pioglitazone 15 (N=130) | Alogliptin 25 + Pioglitazone 15 (N=130) | Placebo + Pioglitazone 30 (N=129) | Alogliptin 12.5 + Pioglitazone 30 (N=130) | Alogliptin 25 + Pioglitazone 30 (N=130) | Placebo + Pioglitazone 45 (N=129) | Alogliptin 12.5 + Pioglitazone 45 (N=130) | Alogliptin 25 + Pioglitazone 45 (N=130)
Headache (Nervous system disorders) | 6 | 5 | 9 | 16 | 5 | 3 | 2 | 2 | 5 | 5 | 6 | 6
Urinary tract infection (Infections and infestations) | 6 | 6 | 5 | 7 | 5 | 6 | 8 | 4 | 4 | 8 | 5 | 5
Nasopharyngitis (Infections and infestations) | 5 | 5 | 4 | 3 | 8 | 8 | 4 | 5 | 9 | 4 | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 7 | 5 | 6 | 5 | 3 | 2 | 8 | 4 | 12 | 3
Diarrhoea (Gastrointestinal disorders) | 11 | 2 | 4 | 5 | 3 | 6 | 4 | 2 | 7 | 5 | 4 | 7
Influenza (Infections and infestations) | 3 | 4 | 4 | 9 | 4 | 8 | 7 | 2 | 8 | 5 | 3 | 2
Dizziness (Nervous system disorders) | 4 | 3 | 2 | 5 | 7 | 2 | 4 | 5 | 5 | 6 | 6 | 1
Hypertension (Vascular disorders) | 4 | 6 | 4 | 6 | 9 | 3 | 2 | 3 | 3 | 2 | 5 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 8 | 3 | 2 | 4 | 1 | 5 | 4 | 2 | 4 | 4
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 7 | 6 | 5 | 2 | 3 | 5 | 2 | 4 | 3 | 3 | 1
Oedema peripheral (General disorders) | 2 | 2 | 2 | 2 | 2 | 7 | 6 | 4 | 1 | 2 | 4 | 6
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 2 | 2 | 2 | 3 | 3 | 7 | 0 | 3 | 5
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 3 | 3 | 1 | 2 | 1 | 4 | 7 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 7 | 0 | 1 | 2 | 1 | 1 | 3 | 1 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.